CLINICAL TRIAL: NCT00985088
Title: A Study to Evaluate the Safety and Immunogenicity of A/California/7/2009 (H1N1)V-like Vaccines GSK2340273A and GSK2340274A in Adults Aged 18 Years and Older
Brief Title: Safety and Immunogenicity of H1N1 Vaccines in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113440
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Influenza
Keywords: GSK Bio's influenza vaccine GSK2340274A; influenza infection; GSK Bio's influenza vaccine GSK2340273A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (8):
- GSK2340274A F1_2D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received 2 doses of Formulation 1 (F1) of GSK2340274A vaccine: at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340274A
- GSK2340274A F2_2D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received 2 doses of Formulation 2 (F2) of GSK2340274A vaccine: at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340274A
- GSK2340274A F2_1D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 2 (F2) of GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and one dose of saline placebo at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340274A; Biological: Saline placebo
- GSK2340274A F1_1D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 1 (F1) of GSK2340274A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and one dose of saline placebo at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340274A; Biological: Saline placebo
- GSK2340273A F1_1D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 1 (F1) of GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and one dose of saline at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340273A; Biological: Saline placebo
- GSK2340273A F2_2D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received 2 doses of Formulation 2 (F2) of GSK2340273A vaccine: at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340273A
- GSK2340273A F2_1D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 2 (F2) of GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and one dose of saline at Day 21, administered intramuscularly into the deltoid region of the dominant arm. Subjects above (>) 60 years old received an additional dose of Formulation 2 (F2) of GSK2340273A vaccine after Day 42, administered into the deltoid region of the non-dominant arm.
  Interventions: Biological: GSK2340273A; Biological: Saline placebo
- GSK2340273A F3_2D Group (Experimental): Healthy male or female subjects, above and including 18 years of age, who received 2 doses of Formulation 3 of GSK2340273A vaccine: at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
  Interventions: Biological: GSK2340273A

INTERVENTIONS:
Biological: GSK2340274A — one or two intramuscular injections
  Arms: GSK2340274A F1_1D Group; GSK2340274A F1_2D Group; GSK2340274A F2_1D Group; GSK2340274A F2_2D Group
Biological: GSK2340273A — one or two intramuscular injections
  Arms: GSK2340273A F1_1D Group; GSK2340273A F2_1D Group; GSK2340273A F2_2D Group; GSK2340273A F3_2D Group
Biological: Saline placebo — One injection
  Arms: GSK2340273A F1_1D Group; GSK2340273A F2_1D Group; GSK2340274A F1_1D Group; GSK2340274A F2_1D Group

SUMMARY:
The purpose of this study is to characterize the safety and immunogenicity of the H1N1 (swine) flu vaccines GSK2340273A and GSK2340274A in adults 18 years of age or older.

This protocol posting has been updated for sections impacted by the Protocol amendment 1, Sept 2009.

DETAILED DESCRIPTION:
Collaborators: United States Department of Health and Human Services, Office of Biomedical Advanced Research and Development Authority

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Male and female adults, >= 18 years of age at the time of the first vaccination.
* Safety laboratory test results within the parameters specified in the protocol.
* Satisfactory baseline medical assessment by history and physical examination.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits as documented by signature on the informed consent document.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of first vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus
* Previous vaccination at any time with an H1N1v-like virus vaccine or a medical history of physician-confirmed infection with an H1N1v-like virus.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC (>=100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination, are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine
* With the exception of seasonal influenza vaccination, administration of any vaccine(s) within 30 days before study vaccination on Day 0. Seasonal influenza vaccine may be administered up to 14 days prior to study vaccination on Day 0.
* Planned administration of any vaccine not foreseen by the study protocol between Day 0 and the Day 42 phlebotomy, including seasonal influenza vaccine or a monovalent pandemic H1N1 vaccine other than the study vaccines.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to the first vaccination.
* Lactating or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1343 (Actual)
Dates: Start 2009-10-11 (Actual); Primary Completion 2009-11-09 (Actual); Study Completion 2010-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (10):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cleveland, Ohio
- Canada (4):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Pointe-Claire, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ferguson M, Risi G, Davis M, Sheldon E, Baron M, Li P, Madariaga M, Fries L, Godeaux O, Vaughn D. Safety and long-term humoral immune response in adults after vaccination with an H1N1 2009 pandemic influenza vaccine with or without AS03 adjuvant. J Infect Dis. 2012 Mar 1;205(5):733-44. doi: 10.1093/infdis/jir641. PMID 22315336
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1343 subjects enrolled in the study, 3 subjects did not receive any vaccination.
Groups:
- GSK2340273A F1_1D Group: Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 1 (F1) of GSK2340273A vaccine at Day 0, administrated intramuscularly into the deltoid region of the non-dominant arm and one dose of saline at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
Period: Overall Study
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Started | 222 | 114 | 112 | 221 | 223 | 115 | 111 | 222
Completed | 211 | 112 | 108 | 214 | 214 | 108 | 107 | 216
Not Completed | 11 | 2 | 4 | 7 | 9 | 7 | 4 | 6
Not completed — Serious Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 1 | 3 | 2 | 1 | 2
Not completed — Migrated/moved from study area | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 6 | 1 | 2 | 6 | 6 | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group | Total
Number analyzed (Participants) | 222 | 114 | 112 | 221 | 223 | 115 | 111 | 222 | 1340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (17.37) | 58.8 (18.69) | 59.3 (17.71) | 58.6 (17.91) | 58.7 (17.59) | 58.4 (17.96) | 58.8 (17.55) | 58.7 (18.16) | 58.7 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 69 | 69 | 138 | 132 | 70 | 75 | 128 | 816
  Male | 87 | 45 | 43 | 83 | 91 | 45 | 36 | 94 | 524
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/ African American | 14 | 7 | 7 | 14 | 9 | 8 | 4 | 12 | 75
  Geographic ancestry: American Indian or Alaskan Native | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 4
  Geographic ancestry: Asian - Central/South Asian heritage | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 3 | 9
  Geographic ancestry: Asian - East Asian heritage | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 6
  Geographic ancestry: Asian - Japanese heritage | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Geographic ancestry: Asian - South East Asian heritage | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 5
  Geographic ancestry: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Geographic ancestry: White - Arabic/North African heritage | 3 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 11
  Geographic ancestry: White - Caucasian/European heritage | 201 | 102 | 101 | 192 | 199 | 98 | 102 | 196 | 1191
  Geographic ancestry: Other | 3 | 1 | 2 | 9 | 10 | 2 | 3 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seropositive for Haemagglutination Inhibition (HI) Antibodies Against the A/California Virus Strain
Description: A seropositive subject against the A/California/ virus strain was defined as a subject with H1N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (≥) the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 60 years (y) old and subjects older than (>) 60 years.
Time Frame: At Day 0
Population: The analysis was performed only on subjects receiving F1 or F2 of GSK2340274A vaccine from the According-to-Protocol (ATP) cohort for immunogenicity, which included all subjects who received the vaccine/placebo doses on Days 0, 21 and for whom assay results for antibodies against A/California-like HA antigen for blood samples taken were available.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340274A F1 Group: Pooled group comprising the subjects from GSK2340274A F1_2D Group and GSK2340274A F1_1D Group.
- GSK2340274A F2 Group: Pooled group comprising the subjects from GSK2340274A F2_1D Group and GSK2340274A F2_2D Group.
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Participants
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 91 | 48
  > 60y | 168 | 75

2. Primary Outcome: Number of Subjects Seropositive for Haemagglutination Inhibition (HI) Antibodies Against the A/California Virus Strain
Description: A seropositive subject against the A/California/ virus strain was defined as a subject with H1N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (≥) the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 60 years (y) old and subjects > 60 years.
Time Frame: At Day 21
Population: The analysis was performed only on subjects receiving F1 or F2 of GSK2340274A vaccine from the ATP cohort for immunogenicity, which included all subjects who received the vaccine/placebo doses on both Days 0 and 21 and for whom assay results for antibodies against A/California-like HA antigen for blood samples taken were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Participants
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 163 | 83
  > 60y | 275 | 136

3. Primary Outcome: Number of Subjects Seropositive for (HI) Antibodies Against the A/California Virus Strain
Description: A seropositive subject against the A/California/ virus strain was defined as a subject with H1N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (≥) the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 64 years (y) old and subjects > 64 years.
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Participants
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 99 | 52
  > 64y | 160 | 71

4. Primary Outcome: Number of Subjects Seropositive for (HI) Antibodies Against the A/California Virus Strain
Description: as for outcome 3
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Participants
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 181 | 93
  > 64y | 257 | 126

5. Primary Outcome: Number of Seroconverted (SCR) Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California Virus Strain
Description: A seroconverted subject was defined as a vaccinated subject who had a post-vaccination titer ≥ 1:40 and at least a 4-fold increase in pre-vaccination titer. The Flu strain assessed was A/California/7/09 (H1N1)v-like) and results were tabulated for subjects between 18 and 60 years of age and older (>60y).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Participants
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 149 | 69
  > 60y | 215 | 82

6. Primary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against A/California Strain
Description: A seroconverted subject was defined as a vaccinated subject who had a post-vaccination titer ≥ 1:40 and at least a 4-fold increase in pre-vaccination titer. The Flu strain assessed was A/California/7/09 (H1N1)v-like) and results were tabulated for subjects between 18 and 64 years and older (>64y).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Participants
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 163 | 75
  > 64y | 201 | 76

7. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The Flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09) and results were tabulated for subjects between 18 and 60 years and older (>60y).
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Participants
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 35 | 17
  > 60y | 35 | 22

8. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The Flu strain assessed was Flu A/CAL/7/09 and results were tabulated for subjects between 18 and 60 years and older (>60y).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Participants
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 160 | 78
  > 60y | 250 | 104

9. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40. The Flu strain assessed was Flu A/CAL/7/09 and results were tabulated for subjects between 18 and 64 years and older (>64y).
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Participants
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 36 | 19
  > 64y | 34 | 20

10. Primary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Strain
Description: as for outcome 9
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Participants
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 176 | 86
  > 64y | 234 | 96

11. Primary Outcome: Seroconversion Factor (SCF) for Haemagglutination Inhibition (HI) Antibodies Against A/California Virus Strain
Description: SCF was defined as the fold increase in serum HI geometric mean ratio (mean[log10(POST/PRE)]) vaccination compared to Day 21. The flu strain assessed was Flu A/CAL/7/09 and results were tabulated for subjects between 18 and 60 years of age and older (>60y).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 275 | 138
Fold increase
  18 - 60y: number analyzed (Participants) | 163 | 83
  18 - 60y | 30.1 [24.5 to 36.9] | 18.5 [13.8 to 24.6]
  > 60y | 10.8 [9.4 to 12.5] | 7.4 [6.0 to 9.2]

12. Primary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against A/California Strain
Description: SCF was defined as the fold increase in serum HI geometric mean ratio (mean[log10(POST/PRE)]) vaccination compared to Day 21. The flu strain assessed was Flu A/CAL/7/09 and results were tabulated for subjects between 18 and 64 years of age and older (>64y).
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A F1 Group | GSK2340274A F2 Group
Number analyzed (Participants) | 257 | 128
Fold increase
  18 - 64y: number analyzed (Participants) | 181 | 93
  18 - 64y | 29.2 [24.0 to 35.6] | 17.0 [13.0 to 22.3]
  > 64y | 10.3 [8.9 to 11.9] | 7.3 [5.9 to 9.2]

13. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against A/California Virus Strain
Description: A seropositive subject against the A/California/ virus strain was defined as a subject with H1N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (≥) the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 60 years (y) old and > 60 years and subjects between 18 and 64 years old and > 64 years, respectively.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all subjects who received the vaccine/ placebo doses on both Days 0 and 21 and from whom assay results for antibodies against A/California-like HA antigen for blood samples taken were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 140 | 70 | 68 | 135 | 137 | 64 | 67 | 136
Participants
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60 y), Day 0 | 47 | 25 | 23 | 44 | 52 | 21 | 22 | 37
  A/California strain (18-60 y), Day 21: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60 y), Day 21 | 80 | 41 | 42 | 83 | 79 | 44 | 43 | 77
  A/California strain (>60 y), Day 0 | 92 | 36 | 39 | 76 | 76 | 30 | 41 | 83
  A/California strain (>60 y), Day 21 | 140 | 68 | 68 | 135 | 129 | 58 | 62 | 124
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64 y), Day 0 | 55 | 28 | 24 | 44 | 57 | 23 | 25 | 40
  A/California strain (18-64 y), Day 21: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64 y), Day 21 | 92 | 46 | 47 | 89 | 88 | 46 | 47 | 86
  A/California strain (>64 y), Day 0: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (>64 y), Day 0 | 84 | 33 | 38 | 76 | 71 | 28 | 38 | 80
  A/California strain (>64 y), Day 21: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (>64 y), Day 21 | 128 | 63 | 63 | 129 | 120 | 56 | 58 | 115

14. Secondary Outcome: Titers for HI Antibodies Against A/California Strain
Description: Antibody titers were presented as geometric mean titers (GMTs), for the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 60 years (y) old and > 60 years and subjects between 18 and 64 years old and > 64 years, respectively.
Time Frame: At Days 0 and 21
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 140 | 70 | 68 | 135 | 137 | 64 | 67 | 136
Titers
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60 y), Day 0 | 13.9 [10.9 to 17.7] | 14.9 [10.1 to 21.8] | 11.3 [8.5 to 14.9] | 12.9 [9.9 to 16.9] | 15.0 [11.7 to 19.2] | 10.6 [7.5 to 14.8] | 11.0 [8.0 to 15.1] | 11.0 [8.6 to 14.1]
  A/California strain (18-60 y), Day 21: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60 y), Day 21 | 415.0 [328.6 to 524.0] | 299.1 [214.6 to 416.9] | 191.7 [139.5 to 263.5] | 391.0 [311.0 to 491.6] | 149.9 [114.0 to 197.2] | 167.6 [113.8 to 246.8] | 231.9 [158.4 to 339.6] | 100.3 [73.3 to 137.5]
  A/California strain (>60 y), Day 0 | 12.8 [11.0 to 15.0] | 10.2 [8.2 to 12.6] | 13.4 [9.9 to 18.0] | 11.9 [10.0 to 14.2] | 11.9 [10.1 to 14.2] | 9.9 [7.7 to 12.7] | 12.4 [9.9 to 15.6] | 12.3 [10.5 to 14.5]
  A/California strain (>60 y), Day 21 | 150.7 [124.1 to 183.1] | 84.1 [62.4 to 113.4] | 88.9 [66.5 to 118.9] | 118.5 [98.3 to 142.9] | 72.6 [57.3 to 92.0] | 47.0 [32.1 to 68.8] | 47.6 [35.0 to 64.9] | 47.3 [36.9 to 60.6]
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64 y), Day 0 | 13.5 [10.8 to 16.8] | 14.5 [10.1 to 20.6] | 10.9 [8.3 to 14.3] | 12.1 [9.4 to 15.6] | 14.5 [11.5 to 18.2] | 11.2 [8.0 to 15.6] | 11.3 [8.4 to 15.3] | 10.8 [8.6 to 13.6]
  A/California strain (18-64 y), Day 21: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64 y), Day 21 | 389.2 [310.9 to 487.3] | 265.2 [191.7 to 366.8] | 172.1 [126.3 to 234.5] | 359.6 [282.1 to 458.3] | 149.1 [114.7 to 193.8] | 183.1 [124.0 to 270.4] | 234.9 [164.4 to 335.7] | 96.6 [72.1 to 129.5]
  A/California strain (>64 y), Day 0: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (>64 y), Day 0 | 13.0 [11.0 to 15.3] | 10.1 [8.1 to 12.6] | 13.9 [10.1 to 19.0] | 12.4 [10.3 to 14.9] | 12.1 [10.1 to 14.5] | 9.4 [7.3 to 12.1] | 12.2 [9.7 to 15.5] | 12.6 [10.6 to 14.9]
  A/California strain (>64 y), Day 21: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (>64 y), Day 21 | 143.5 [117.5 to 175.4] | 83.0 [60.5 to 113.9] | 90.7 [66.7 to 123.3] | 118.8 [98.8 to 142.9] | 69.3 [54.3 to 88.3] | 42.2 [29.4 to 60.6] | 42.7 [31.5 to 57.8] | 46.0 [35.5 to 59.8]

15. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against A/California Virus Strain
Description: A seroconverted subject was defined as a vaccinated subject who had a post-vaccination titer ≥ 1:40 and at least a 4-fold increase in pre-vaccination titer. The Flu strain assessed was A/California/7/09 (H1N1)v-like) and results were tabulated for subjects between 18-60 years of age and older (>60y) and for subjects between 18-64 years old and >64 years.
Time Frame: At Day 21
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 140 | 70 | 68 | 135 | 137 | 64 | 67 | 136
Participants
  A/California strain, 18-60y: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain, 18-60y | 74 | 34 | 35 | 75 | 58 | 35 | 33 | 49
  A/California strain, > 60y | 109 | 45 | 37 | 106 | 69 | 24 | 27 | 52
  A/California strain, 18-64y: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain, 18-64y | 84 | 38 | 37 | 79 | 64 | 37 | 37 | 55
  A/California strain, > 64y: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain, > 64y | 99 | 41 | 35 | 102 | 63 | 22 | 23 | 46

16. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against HI Antibodies for the A/California Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum HI antibody titers ≥ 1:40. The Flu strain assessed was A/California/7/09 (H1N1)v-like) and results were tabulated for subjects between 18-60 years of age and older (>60y) and for subjects between 18-64 years old and >64 years.
Time Frame: At Days 0 and 21
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 140 | 70 | 68 | 135 | 137 | 64 | 67 | 136
Participants
  A/California strain (18-60y), Day 0: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60y), Day 0 | 18 | 10 | 7 | 17 | 19 | 7 | 6 | 13
  A/California strain (18-60y), Day 21: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain (18-60y), Day 21 | 79 | 40 | 38 | 81 | 71 | 39 | 41 | 61
  A/California strain (> 60y), Day 0 | 16 | 9 | 13 | 19 | 23 | 7 | 12 | 18
  A/California strain (> 60y), Day 21 | 127 | 55 | 49 | 123 | 93 | 32 | 39 | 74
  A/California strain (18-64y), Day 0: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64y), Day 0 | 19 | 11 | 8 | 17 | 20 | 8 | 7 | 14
  A/California strain (18-64y), Day 21: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain (18-64y), Day 21 | 91 | 45 | 41 | 85 | 79 | 41 | 45 | 68
  A/California strain (> 64y), Day 0: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (> 64y), Day 0 | 15 | 8 | 12 | 19 | 22 | 6 | 11 | 17
  A/California strain (> 64y), Day 21: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain (> 64y), Day 21 | 115 | 50 | 46 | 119 | 85 | 30 | 35 | 67

17. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against A/California Virus Strain
Description: SCF was defined as the fold increase in serum HI geometric mean ratio (mean[log10(POST/PRE)]) vaccination compared to Day 21. The flu strain assessed was Flu A/CAL/7/09 and results were tabulated for subjects between 18-60 years of age and older (> 60y) and for subjects between 18-64 years old and > 64 years.
Time Frame: At Day 21
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 140 | 70 | 68 | 135 | 137 | 64 | 67 | 136
Fold increase
  A/California strain, 18-60y: number analyzed (Participants) | 80 | 41 | 42 | 83 | 80 | 44 | 43 | 82
  A/California strain, 18-60y | 29.9 [22.4 to 40.0] | 20.1 [13.0 to 31.2] | 17.0 [11.4 to 25.2] | 30.2 [22.4 to 40.7] | 10.0 [7.3 to 13.6] | 15.9 [10.4 to 24.2] | 21.1 [12.9 to 34.5] | 9.1 [6.6 to 12.7]
  A/California strain, > 60y | 11.8 [9.6 to 14.4] | 8.3 [6.0 to 11.3] | 6.7 [5.0 to 8.9] | 9.9 [8.1 to 12.1] | 6.1 [4.9 to 7.6] | 4.8 [3.3 to 6.8] | 3.8 [2.9 to 5.1] | 3.8 [3.1 to 4.8]
  A/California strain, 18-64y: number analyzed (Participants) | 92 | 46 | 47 | 89 | 89 | 46 | 47 | 91
  A/California strain, 18-64y | 28.8 [22.0 to 37.9] | 18.3 [12.1 to 27.8] | 15.8 [11.0 to 22.7] | 29.6 [22.1 to 39.8] | 10.3 [7.7 to 13.8] | 16.4 [10.9 to 24.5] | 20.7 [13.0 to 33.0] | 8.9 [6.6 to 12.2]
  A/California strain, > 64y: number analyzed (Participants) | 128 | 65 | 63 | 129 | 128 | 62 | 63 | 127
  A/California strain, > 64y | 11.1 [9.0 to 13.6] | 8.2 [6.0 to 11.4] | 6.5 [4.8 to 8.9] | 9.6 [7.9 to 11.6] | 5.7 [4.6 to 7.2] | 4.5 [3.1 to 6.4] | 3.5 [2.7 to 4.6] | 3.7 [2.9 to 4.6]

18. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against the A/California Virus Strain
Description: A seropositive subject against the A/California/ virus strain was defined as a subject with H1N1 reciprocal HI antibody titers greater than or equal to (≥) the seropositivity cut-off of 1:10. Results were tabulated according to age strata: subjects between 18 to 60 years (y) old and > 60 years and subjects between 18 and 64 years old and > 64 years, respectively.
Time Frame: At Days 0 and 42
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 64 | 69 | 68 | 67 | 64 | 64 | 63 | 69
Participants
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain (18-60 y), Day 0 | 24 | 24 | 21 | 23 | 26 | 20 | 22 | 15
  A/California strain (18-60 y), Day 42: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain (18-60 y), Day 42 | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 37
  A/California strain (> 60 y), Day 0 | 39 | 36 | 39 | 42 | 33 | 31 | 40 | 44
  A/California strain (> 60 y), Day 42 | 64 | 68 | 68 | 67 | 59 | 61 | 56 | 68
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain (18-64 y), Day 0 | 25 | 27 | 22 | 23 | 28 | 22 | 25 | 16
  A/California strain (18-64 y), Day 42: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain (18-64 y), Day 42 | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 41
  A/California strain (> 64 y), Day 0: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain (> 64 y), Day 0 | 38 | 33 | 38 | 42 | 31 | 29 | 37 | 43
  A/California strain (> 64 y), Day 42: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain (> 64 y), Day 42 | 61 | 63 | 63 | 63 | 56 | 59 | 52 | 64

19. Secondary Outcome: Titers for HI Antibodies Against the A/California Virus Strain
Description: as for outcome 14
Time Frame: At Days 0 and 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 64 | 69 | 68 | 67 | 64 | 64 | 63 | 69
Titers
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain (18-60 y), Day 0 | 14.8 [10.1 to 21.5] | 14.3 [9.8 to 20.7] | 10.9 [8.2 to 14.5] | 13.4 [9.3 to 19.3] | 15.2 [10.8 to 21.4] | 10.6 [7.5 to 14.9] | 11.0 [8.0 to 15.1] | 9.5 [6.8 to 13.1]
  A/California strain (18-60 y), Day 42: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain (18-60 y), Day 42 | 565.0 [447.1 to 714.1] | 468.9 [351.1 to 626.1] | 139.2 [100.6 to 192.7] | 301.1 [206.4 to 439.2] | 99.9 [65.2 to 153.1] | 197.4 [142.1 to 274.1] | 203.8 [140.6 to 295.4] | 84.3 [55.1 to 128.8]
  A/California strain (> 60 y), Day 0 | 11.2 [9.1 to 13.8] | 10.3 [8.3 to 12.8] | 13.4 [9.9 to 18.0] | 13.5 [10.5 to 17.3] | 10.8 [8.6 to 13.6] | 10.0 [7.8 to 12.8] | 12.9 [10.2 to 16.4] | 11.4 [9.4 to 13.9]
  A/California strain (> 60 y), Day 42 | 235.1 [178.2 to 310.2] | 146.1 [107.4 to 198.6] | 76.8 [57.9 to 101.8] | 108.6 [83.0 to 142.1] | 65.1 [46.5 to 91.2] | 55.9 [39.3 to 79.4] | 41.8 [30.1 to 58.0] | 58.2 [43.2 to 78.4]
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain (18-64 y), Day 0 | 14.2 [9.9 to 20.4] | 13.9 [9.9 to 19.6] | 10.5 [8.0 to 13.9] | 12.3 [8.7 to 17.2] | 15.0 [10.8 to 20.8] | 11.2 [8.0 to 15.7] | 11.3 [8.4 to 15.3] | 9.4 [6.9 to 12.9]
  A/California strain (18-64 y), Day 42: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain (18-64 y), Day 42 | 503.9 [386.3 to 657.4] | 424.9 [319.5 to 565.0] | 125.0 [91.2 to 171.2] | 254.6 [171.8 to 377.2] | 97.6 [65.5 to 145.3] | 214.5 [153.5 to 299.6] | 210.2 [147.5 to 299.6] | 81.9 [55.7 to 120.4]
  A/California strain (> 64 y), Day 0: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain (> 64 y), Day 0 | 11.3 [9.1 to 14.0] | 10.2 [8.2 to 12.7] | 13.9 [10.1 to 19.0] | 14.3 [11.1 to 18.6] | 10.7 [8.5 to 13.6] | 9.5 [7.4 to 12.3] | 12.8 [10.0 to 16.4] | 11.6 [9.5 to 14.1]
  A/California strain (> 64 y), Day 42: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain (> 64 y), Day 42 | 243.7 [183.7 to 323.2] | 142.7 [103.1 to 197.5] | 79.1 [58.8 to 106.6] | 114.4 [87.2 to 150.2] | 64.8 [45.5 to 92.2] | 50.5 [36.2 to 70.4] | 36.6 [26.8 to 50.0] | 58.0 [42.3 to 79.6]

20. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against A/California Virus Strain
Description: as for outcome 15
Time Frame: At Day 42
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 64 | 69 | 68 | 67 | 64 | 64 | 63 | 69
Participants
  A/California strain, 18-60 y: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain, 18-60 y | 36 | 37 | 31 | 37 | 21 | 38 | 32 | 25
  A/California strain, > 60 y | 54 | 54 | 37 | 50 | 38 | 30 | 22 | 36
  A/California strain, 18-64 y: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain, 18-64 y | 38 | 41 | 33 | 39 | 23 | 40 | 36 | 28
  A/California strain, > 64 y: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain, > 64 y | 52 | 50 | 35 | 48 | 36 | 28 | 18 | 33

21. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Strain
Description: as for outcome 16
Time Frame: At Days 0 and 42
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 64 | 69 | 68 | 67 | 64 | 64 | 63 | 69
Participants
  A/California (18-60 y), Day 0: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California (18-60 y), Day 0 | 10 | 9 | 6 | 9 | 9 | 7 | 6 | 4
  A/California (18-60 y), Day 42: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California (18-60 y), Day 42 | 39 | 39 | 35 | 38 | 32 | 42 | 40 | 30
  A/California (> 60 y), Day 0 | 3 | 9 | 13 | 11 | 11 | 7 | 12 | 7
  A/California (> 60 y), Day 42 | 62 | 60 | 50 | 58 | 46 | 39 | 36 | 44
  A/California (18-64 y), Day 0: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California (18-64 y), Day 0 | 10 | 10 | 7 | 9 | 10 | 8 | 7 | 5
  A/California (18-64 y), Day 42: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California (18-64 y), Day 42 | 42 | 44 | 38 | 40 | 35 | 44 | 44 | 34
  A/California (> 64 y), Day 0: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California (> 64 y), Day 0 | 3 | 8 | 12 | 11 | 10 | 6 | 11 | 6
  A/California (> 64 y), Day 42: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California (> 64 y), Day 42 | 59 | 55 | 47 | 56 | 43 | 37 | 32 | 40

22. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against A/California Virus Strain
Description: as for outcome 17
Time Frame: At Day 42
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 64 | 69 | 68 | 67 | 64 | 64 | 63 | 69
Fold increase
  A/California strain, 18-60 y: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 43 | 43 | 39
  A/California strain, 18-60 y | 38.3 [25.6 to 57.2] | 32.9 [21.2 to 51.0] | 12.8 [8.7 to 18.8] | 22.4 [15.0 to 33.6] | 6.6 [4.1 to 10.6] | 18.7 [12.7 to 27.4] | 18.5 [11.5 to 29.7] | 8.9 [5.7 to 13.8]
  A/California strain, > 60 y | 21.1 [14.8 to 29.9] | 14.2 [10.2 to 19.7] | 5.8 [4.4 to 7.6] | 8.1 [6.2 to 10.4] | 6.0 [4.3 to 8.5] | 5.6 [4.0 to 7.7] | 3.2 [2.4 to 4.3] | 5.1 [3.8 to 6.8]
  A/California strain, 18-64 y: number analyzed (Participants) | 42 | 44 | 45 | 44 | 42 | 45 | 47 | 43
  A/California strain, 18-64 y | 35.4 [23.6 to 53.1] | 30.5 [20.0 to 46.6] | 11.9 [8.4 to 16.8] | 20.8 [14.1 to 30.6] | 6.5 [4.2 to 10.2] | 19.1 [13.2 to 27.6] | 18.6 [11.9 to 28.9] | 8.7 [5.8 to 13.1]
  A/California strain, > 64 y: number analyzed (Participants) | 61 | 64 | 63 | 63 | 61 | 62 | 59 | 65
  A/California strain, > 64 y | 21.6 [15.1 to 30.8] | 14.0 [9.9 to 19.7] | 5.7 [4.2 to 7.7] | 8.0 [6.1 to 10.4] | 6.0 [4.2 to 8.6] | 5.3 [3.8 to 7.3] | 2.9 [2.2 to 3.7] | 5.0 [3.7 to 6.8]

23. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against the A/California Virus Strain
Description: as for outcome 18
Time Frame: At Days 0 and 182
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 136 | 66 | 67 | 134 | 132 | 64 | 63 | 137
Participants
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 0 | 46 | 25 | 23 | 44 | 50 | 20 | 20 | 35
  A/California strain (18-60 y), Day 182: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 182 | 75 | 42 | 40 | 79 | 72 | 43 | 40 | 76
  A/California strain (> 60 y), Day 0 | 89 | 33 | 39 | 76 | 73 | 31 | 41 | 82
  A/California strain (> 60 y), Day 182 | 136 | 66 | 60 | 133 | 114 | 52 | 54 | 116
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 0 | 54 | 28 | 24 | 44 | 55 | 22 | 23 | 38
  A/California strain (18-64 y), Day 182: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 182 | 87 | 47 | 44 | 85 | 81 | 45 | 44 | 84
  A/California strain (> 64 y), Day 0: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (> 64 y), Day 0 | 81 | 30 | 38 | 76 | 68 | 29 | 38 | 79
  A/California strain (> 64 y), Day 182: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (> 64 y), Day 182 | 124 | 61 | 56 | 127 | 105 | 50 | 50 | 108

24. Secondary Outcome: Titers for HI Antibodies Against the A/California Virus Strain
Description: as for outcome 14
Time Frame: At Days 0 and 182
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 136 | 66 | 67 | 134 | 132 | 64 | 63 | 137
Titers
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 0 | 14.5 [11.3 to 18.6] | 14.5 [9.9 to 21.1] | 11.5 [8.7 to 15.3] | 13.4 [10.2 to 17.6] | 15.1 [11.7 to 19.4] | 10.2 [7.3 to 14.3] | 10.8 [7.7 to 15.1] | 10.4 [8.3 to 13.1]
  A/California strain (18-60 y), Day 182: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 182 | 250.3 [195.0 to 321.3] | 184.1 [130.7 to 259.3] | 77.9 [55.3 to 109.8] | 149.2 [113.9 to 195.4] | 92.1 [67.9 to 124.9] | 92.4 [65.1 to 131.3] | 133.3 [89.9 to 197.7] | 66.6 [50.9 to 87.2]
  A/California strain (>60 y), Day 0 | 12.6 [10.8 to 14.8] | 10.3 [8.2 to 12.9] | 13.5 [10.0 to 18.3] | 11.9 [9.9 to 14.2] | 12.1 [10.1 to 14.4] | 10.0 [7.8 to 12.8] | 13.2 [10.4 to 16.7] | 12.1 [10.3 to 14.2]
  A/California strain (>60 y), Day 182 | 106.6 [87.9 to 129.2] | 59.2 [44.2 to 79.5] | 37.9 [27.3 to 52.6] | 49.7 [41.2 to 59.8] | 42.5 [33.6 to 53.7] | 34.9 [24.2 to 50.4] | 38.7 [27.4 to 54.6] | 34.2 [27.3 to 42.7]
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 0 | 14.0 [11.2 to 17.6] | 14.1 [10.0 to 20.0] | 11.1 [8.5 to 14.6] | 12.5 [9.7 to 16.2] | 14.5 [11.5 to 18.3] | 10.9 [7.8 to 15.2] | 11.2 [8.1 to 15.3] | 10.3 [8.3 to 12.8]
  A/California strain (18-64 y), Day 182: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 182 | 232.7 [183.5 to 295.0] | 166.0 [118.2 to 233.1] | 65.7 [46.1 to 93.6] | 132.3 [100.6 to 174.0] | 90.7 [68.5 to 120.0] | 100.7 [70.6 to 143.8] | 138.8 [96.2 to 200.2] | 63.0 [48.7 to 81.4]
  A/California strain (>64 y), Day 0: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (>64 y), Day 0 | 12.8 [10.8 to 15.1] | 10.2 [8.0 to 12.8] | 14.1 [10.3 to 19.4] | 12.4 [10.3 to 14.8] | 12.2 [10.1 to 14.7] | 9.5 [7.4 to 12.3] | 13.0 [10.2 to 16.6] | 12.3 [10.4 to 14.6]
  A/California strain (>64 y), Day 182: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (>64 y), Day 182 | 103.3 [84.6 to 126.3] | 58.5 [43.1 to 79.3] | 40.6 [28.9 to 57.0] | 51.1 [42.3 to 61.8] | 40.5 [31.7 to 51.8] | 31.8 [22.3 to 45.3] | 34.5 [24.5 to 48.7] | 33.9 [26.8 to 42.8]

25. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies
Description: as for outcome 15
Time Frame: At Day 182
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 136 | 66 | 67 | 134 | 132 | 64 | 63 | 137
Participants
  A/California strain, 18-60 y: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain, 18-60 y | 71 | 36 | 26 | 57 | 44 | 29 | 28 | 45
  A/California strain, > 60 y | 93 | 34 | 16 | 55 | 52 | 25 | 21 | 40
  A/California strain, 18-64 y: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain, 18-64 y | 79 | 38 | 26 | 59 | 50 | 31 | 32 | 46
  A/California strain, > 64 y: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain, > 64 y | 85 | 32 | 16 | 53 | 46 | 23 | 17 | 39

26. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against A/California Virus Strain
Description: as for outcome 16
Time Frame: At Days 0 and 182
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 136 | 66 | 67 | 134 | 132 | 64 | 63 | 137
Participants
  A/California strain (18-60 y), Day 0: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 0 | 18 | 10 | 7 | 17 | 17 | 6 | 6 | 12
  A/California strain (18-60 y), Day 182: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain (18-60 y), Day 182 | 75 | 39 | 33 | 70 | 58 | 35 | 33 | 57
  A/California strain (> 60 y), Day 0 | 15 | 9 | 13 | 18 | 23 | 7 | 12 | 18
  A/California strain (> 60 y), Day 182 | 109 | 44 | 32 | 85 | 75 | 31 | 33 | 69
  A/California strain (18-64 y), Day 0: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 0 | 19 | 11 | 8 | 17 | 18 | 7 | 7 | 13
  A/California strain (18-64 y), Day 182: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain (18-64 y), Day 182 | 85 | 42 | 34 | 72 | 65 | 37 | 37 | 61
  A/California strain (> 64 y), Day 0: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (> 64 y), Day 0 | 14 | 8 | 12 | 18 | 22 | 6 | 11 | 17
  A/California strain (> 64 y), Day 182: number analyzed (Participants) | 124 | 61 | 62 | 128 | 123 | 62 | 59 | 128
  A/California strain (> 64 y), Day 182 | 99 | 41 | 31 | 83 | 68 | 29 | 29 | 65

27. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Against A/California Virus Strain
Description: as for outcome 17
Time Frame: At Day 182
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 136 | 66 | 67 | 134 | 132 | 64 | 63 | 137
Fold increase
  A/California strain, 18-60 y: number analyzed (Participants) | 76 | 42 | 41 | 80 | 76 | 43 | 40 | 80
  A/California strain, 18-60 y | 17.2 [12.8 to 23.3] | 12.7 [8.5 to 19.1] | 6.8 [4.7 to 9.8] | 11.1 [8.2 to 15.1] | 6.1 [4.4 to 8.5] | 9.0 [6.1 to 13.4] | 12.3 [7.5 to 20.4] | 6.4 [4.8 to 8.5]
  A/California strain, > 60 y | 8.4 [6.9 to 10.3] | 5.8 [4.3 to 7.7] | 2.8 [2.1 to 3.7] | 4.2 [3.5 to 5.0] | 3.5 [2.8 to 4.4] | 3.5 [2.5 to 4.9] | 2.9 [2.3 to 3.8] | 2.8 [2.4 to 3.4]
  A/California strain, 18-64 y: number analyzed (Participants) | 88 | 47 | 46 | 86 | 85 | 45 | 44 | 89
  A/California strain, 18-64 y | 16.6 [12.6 to 21.9] | 11.7 [7.9 to 17.5] | 5.9 [4.2 to 8.4] | 10.6 [7.9 to 14.1] | 6.3 [4.6 to 8.5] | 9.3 [6.3 to 13.6] | 12.4 [7.8 to 19.8] | 6.1 [4.7 to 8.0]
  A/California strain, > 64 y: number analyzed (Participants) | 124 | 61 | 62 | 134 | 123 | 62 | 59 | 128
  A/California strain, > 64 y | 8.1 [6.5 to 10.0] | 5.8 [4.3 to 7.7] | 2.9 [2.2 to 3.8] | 4.1 [3.5 to 5.0] | 3.3 [2.6 to 4.2] | 3.3 [2.4 to 4.6] | 2.7 [2.1 to 3.4] | 2.7 [2.3 to 3.3]

28. Secondary Outcome: Adjusted Geometric Mean Titer (GMT) Ratios of A/California Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled group GSK2340274A F1 and GSK2340273A F3_2D Group.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F1 vaccine versus GSK2340273A F3 vaccine
Measure: Number; unit: Titers
Arm/Group | GSK2340274A F1 Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 275 | 136
Titers
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 163 | 82
  Adjusted A/California ratio, 18-60y | 404.9 | 104.5
  Adjusted A/California ratio, > 60y | 152.7 | 55.0
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 181 | 91
  Adjusted A/California ratio, 18-64y | 381.7 | 101.6
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 257 | 127
  Adjusted A/California ratio, > 64y | 156.0 | 56.2

29. Secondary Outcome: Adjusted Geometric Mean Titer (GMT) Ratios of A/California Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled groups GSK2340274A F1 and GSK2340273A F2.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F1 vaccine versus GSK2340273A F2 vaccine
Measure: Number; unit: Titer
Groups:
- GSK2340273A F2 Group: Pooled group comprising the subjects from GSK2340273A F2_1D Group and GSK2340273A F2_2D Group.
Arm/Group | GSK2340274A F1 Group | GSK2340273A F2 Group
Number analyzed (Participants) | 275 | 131
Titer
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 163 | 87
  Adjusted A/California ratio, 18-60y | 400.8 | 215.3
  Adjusted A/California ratio, > 60y | 162.3 | 61.4
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 181 | 93
  Adjusted A/California ratio, 18-64y | 385.7 | 220.2
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 257 | 125
  Adjusted A/California ratio, > 64y | 159.2 | 56.8

30. Secondary Outcome: Adjusted GMT Ratios of A/California Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled group GSK2340274A F1 and the GSK2340273A F1_1D Group.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F1 vaccine vs GSK2340273A F1_1D vaccine
Measure: Number; unit: Titer
Groups:
- GSK2340273A F1_1D Group: Healthy male or female subjects, above and including 18 years of age, who received one dose of Formulation 1 (F1) of GSK2340273A vaccine at Day 0, administered intramuscularly into the deltoid region of the non-dominant arm and one dose of saline placebo at Day 21, administered intramuscularly into the deltoid region of the dominant arm.
Arm/Group | GSK2340274A F1 Group | GSK2340273A F1_1D Group
Number analyzed (Participants) | 275 | 137
Titer
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 163 | 80
  Adjusted A/California ratio, 18-60y | 414.8 | 153.1
  Adjusted A/California ratio, > 60y | 172.9 | 95.6
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 181 | 89
  Adjusted A/California ratio, 18-64y | 393.8 | 151.6
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 257 | 128
  Adjusted A/California ratio, > 64y | 169.9 | 94.2

31. Secondary Outcome: Adjusted GMT Ratios of A/California Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled group GSK2340274A F2 and the GSK2340273A F3_2D Group.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F2 vaccine versus GSK2340273A F3 vaccine
Measure: Number; unit: Titer
Groups:
- GSK2340274A F2 Group: Pooled group comprising the subjects from GSK2340274A F2_2D Group and GSK2340274A F2_1D Group.
Arm/Group | GSK2340274A F2 Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 138 | 136
Titer
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 83 | 82
  Adjusted A/California ratio, 18-60y | 238.2 | 102.3
  Adjusted A/California ratio, > 60y | 113.3 | 61.3
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 93 | 91
  Adjusted A/California ratio, 18-64y | 213.9 | 99.5
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 128 | 127
  Adjusted A/California ratio, > 64y | 117.2 | 60.5

32. Secondary Outcome: Adjusted GMT Ratios for A/California Virus Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled groups GSK2340274A F2 and GSK2340273A F2.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F2 vaccine versus GSK2340273A F2 vaccine
Measure: Number; unit: Titer
Groups:
- GSK2340273A F2 Group: Pooled group comprising the subjects from GSK2340273A F2_2D Group and GSK2340273A F2_1D Group.
Arm/Group | GSK2340274A F2 Group | GSK2340273A F2 Group
Number analyzed (Participants) | 138 | 131
Titer
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 83 | 87
  Adjusted A/California ratio, 18-60y | 234.3 | 208.6
  Adjusted A/California ratio, > 60y | 119.9 | 68.3
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 93 | 93
  Adjusted A/California ratio, 18-64y | 213.7 | 216.7
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 128 | 125
  Adjusted A/California ratio, > 64y | 118.2 | 61.6

33. Secondary Outcome: Adjusted GMT Ratios for A/California Strain
Description: Titers were presented as geometric mean titers (GMTs). Adjusted GMT was defined as the geometric mean antibody titer adjusted for Previous Vaccination baseline titers and results were tabulated for subjects between 18-60 years, > 60 years, 18-64 years and > 64 years, from the pooled group GSK2340274A F2 and the GSK2340273A F1_1D Group.
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all subjects who received the vaccine/placebo doses on Days 0 and 21 and for whom assay results for antibodies against vaccine antigen for blood samples taken were available. This analysis focused on subjects receiving GSK2340274A F2 vaccine vs. GSK2340273A F1_1D vaccine
Measure: Number; unit: Titer
Arm/Group | GSK2340274A F2 Group | GSK2340273A F1_1D Group
Number analyzed (Participants) | 138 | 137
Titer
  Adjusted A/California ratio, 18-60y: number analyzed (Participants) | 83 | 80
  Adjusted A/California ratio, 18-60y | 246.4 | 150.9
  Adjusted A/California ratio, > 60y | 129.6 | 110.2
  Adjusted A/California ratio, 18-64y: number analyzed (Participants) | 93 | 89
  Adjusted A/California ratio, 18-64y | 221.8 | 150.4
  Adjusted A/California ratio, > 64y: number analyzed (Participants) | 128 | 128
  Adjusted A/California ratio, > 64y | 130.7 | 106.3

34. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses, for subjects between 18-64 years of age
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received at least 1 study vaccination and had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 49 | 47 | 92
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Pain, Dose 1 | 74 | 39 | 35 | 80 | 25 | 10 | 11 | 16
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Pain, Dose 1 | 4 | 3 | 0 | 2 | 0 | 0 | 0 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Redness, Dose 1 | 2 | 0 | 2 | 7 | 0 | 0 | 0 | 3
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Swelling, Dose 1 | 3 | 0 | 1 | 9 | 2 | 0 | 0 | 2
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Pain, Dose 2 | 68 | 37 | 4 | 12 | 15 | 7 | 4 | 10
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Pain, Dose 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Redness, Dose 2 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Swelling, Dose 2 | 5 | 3 | 0 | 0 | 1 | 0 | 0 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 81 | 43 | 36 | 80 | 28 | 15 | 13 | 23
  Grade 3 Pain, Across doses | 6 | 5 | 0 | 2 | 1 | 0 | 0 | 0
  Any Redness, Across doses | 6 | 0 | 2 | 7 | 1 | 0 | 0 | 3
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 7 | 3 | 1 | 9 | 3 | 0 | 0 | 3
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 34
Time Frame: During the 7-day (Day 0-6) post-vaccination period following each dose and across doses, for subjects > 64 years of age
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 64 | 130
Participants
  Any Pain, Dose 1 | 73 | 28 | 21 | 75 | 17 | 4 | 4 | 10
  Grade 3 Pain, Dose 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Redness, Dose 1 | 6 | 0 | 0 | 6 | 1 | 1 | 0 | 2
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 9 | 3 | 3 | 9 | 4 | 2 | 0 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Pain, Dose 2 | 63 | 23 | 1 | 4 | 3 | 6 | 3 | 7
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Pain, Dose 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Redness, Dose 2 | 12 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Swelling, Dose 2 | 8 | 3 | 1 | 3 | 0 | 0 | 0 | 1
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 87 | 33 | 21 | 76 | 19 | 10 | 7 | 15
  Grade 3 Pain, Across doses | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Redness, Across doses | 16 | 0 | 1 | 7 | 1 | 1 | 0 | 2
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 13 | 5 | 3 | 11 | 4 | 2 | 0 | 2
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)], headache, joint pain at other location, muscle aches, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Day 0-6) post-vaccination period following each dose and across doses, for subjects between 18-64 years of age
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 49 | 47 | 92
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Fatigue, Dose 1 | 27 | 15 | 8 | 26 | 24 | 13 | 8 | 20
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Fatigue, Dose 1 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0
  Related Fatigue, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Fatigue, Dose 1 | 27 | 15 | 5 | 21 | 20 | 12 | 5 | 13
  Any Headache, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Headache, Dose 1 | 33 | 13 | 15 | 32 | 26 | 15 | 11 | 27
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Headache, Dose 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Related Headache, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Headache, Dose 1 | 28 | 13 | 8 | 20 | 18 | 11 | 9 | 22
  Any Joint pain at other location, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Joint pain at other location, Dose 1 | 15 | 10 | 5 | 15 | 13 | 4 | 2 | 10
  Grade 3 Joint pain at other location, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Joint pain at other location, Dose 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1
  Related Joint pain at other location, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Joint pain at other location, Dose 1 | 14 | 10 | 2 | 12 | 10 | 3 | 1 | 6
  Any Muscle aches, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Muscle aches, Dose 1 | 32 | 19 | 7 | 33 | 15 | 10 | 4 | 17
  Grade 3 Muscle aches, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Muscle aches, Dose 1 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 0
  Related Muscle aches, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Muscle aches, Dose 1 | 29 | 19 | 6 | 26 | 11 | 8 | 2 | 9
  Any Shivering, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Shivering, Dose 1 | 10 | 7 | 0 | 8 | 9 | 2 | 3 | 9
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Shivering, Dose 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Related Shivering, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Shivering, Dose 1 | 9 | 7 | 0 | 6 | 7 | 2 | 3 | 4
  Any Sweating, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Sweating, Dose 1 | 6 | 3 | 0 | 4 | 7 | 2 | 5 | 8
  Grade 3 Sweating, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Related Sweating, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Sweating, Dose 1 | 5 | 3 | 0 | 3 | 5 | 2 | 3 | 7
  Any Temperature, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Any Temperature, Dose 1 | 3 | 1 | 0 | 1 | 3 | 0 | 3 | 3
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 93 | 46 | 47 | 91 | 92 | 49 | 47 | 92
  Related Temperature, Dose 1 | 2 | 1 | 0 | 1 | 2 | 0 | 2 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Fatigue, Dose 2 | 26 | 16 | 4 | 13 | 15 | 10 | 7 | 15
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Fatigue, Dose 2 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Fatigue, Dose 2 | 22 | 13 | 3 | 11 | 13 | 10 | 6 | 8
  Any Headache, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Headache, Dose 2 | 23 | 15 | 3 | 14 | 22 | 17 | 12 | 18
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Headache, Dose 2 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Headache, Dose 2 | 20 | 12 | 1 | 11 | 15 | 16 | 8 | 13
  Any Joint pain at other location, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Joint pain at other location, Dose 2 | 18 | 6 | 1 | 2 | 9 | 4 | 5 | 6
  Grade 3 Joint pain at other location, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Joint pain at other location, Dose 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Joint pain at other location, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Joint pain at other location, Dose 2 | 18 | 4 | 1 | 2 | 7 | 4 | 5 | 3
  Any Muscle aches, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Muscle aches, Dose 2 | 29 | 13 | 2 | 7 | 12 | 7 | 5 | 13
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Muscle aches, Dose 2 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Muscle aches, Dose 2 | 27 | 12 | 2 | 6 | 10 | 7 | 5 | 8
  Any Shivering, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Shivering, Dose 2 | 13 | 5 | 1 | 3 | 8 | 4 | 0 | 3
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Shivering, Dose 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Shivering, Dose 2 | 11 | 3 | 1 | 2 | 6 | 4 | 0 | 2
  Any Sweating, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Sweating, Dose 2 | 9 | 2 | 0 | 2 | 6 | 0 | 2 | 3
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Sweating, Dose 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Sweating, Dose 2 | 8 | 2 | 0 | 2 | 5 | 0 | 1 | 2
  Any Temperature, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Any Temperature, Dose 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 2
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 93 | 46 | 46 | 90 | 90 | 48 | 47 | 91
  Related Temperature, Dose 2 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Any Fatigue, Across doses | 37 | 24 | 9 | 33 | 30 | 18 | 12 | 25
  Grade 3 Fatigue, Across doses | 5 | 3 | 0 | 1 | 3 | 0 | 0 | 0
  Related Fatigue, Across doses | 35 | 22 | 7 | 26 | 26 | 17 | 9 | 18
  Any Headache, Across doses | 43 | 22 | 15 | 37 | 34 | 23 | 18 | 36
  Grade 3 Headache, Across doses | 4 | 3 | 1 | 0 | 2 | 0 | 0 | 1
  Related Headache, Across doses | 38 | 19 | 8 | 26 | 24 | 22 | 12 | 28
  Any Joint pain at other location, Across doses | 26 | 11 | 5 | 17 | 16 | 7 | 6 | 13
  Grade 3 Joint pain at other location, Across doses | 4 | 0 | 0 | 1 | 2 | 0 | 0 | 1
  Related Joint pain at other location, Across doses | 25 | 11 | 3 | 14 | 12 | 6 | 6 | 8
  Any Muscle aches, Across doses | 42 | 22 | 8 | 34 | 21 | 14 | 8 | 24
  Grade 3 Muscle aches, Across doses | 7 | 4 | 0 | 2 | 1 | 0 | 0 | 0
  Related Muscle aches, Across doses | 40 | 21 | 8 | 27 | 15 | 13 | 7 | 15
  Any Shivering, Across doses | 21 | 8 | 1 | 11 | 12 | 5 | 3 | 11
  Grade 3 Shivering, Across doses | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  Related Shivering, Across doses | 18 | 7 | 1 | 8 | 10 | 5 | 3 | 6
  Any Sweating, Across doses | 14 | 4 | 0 | 6 | 12 | 2 | 6 | 9
  Grade 3 Sweating, Across doses | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Related Sweating, Across doses | 13 | 4 | 0 | 5 | 9 | 2 | 3 | 7
  Any Temperature, Across doses | 6 | 2 | 0 | 2 | 4 | 0 | 3 | 4
  Grade 3 Temperature, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Related Temperature, Across doses | 5 | 2 | 0 | 2 | 2 | 0 | 2 | 0

37. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 36
Time Frame: During the 7-day (Day 0-6) post-vaccination period following each dose and across doses, for subjects > 64 years of age
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 64 | 130
Participants
  Any Fatigue, Dose 1 | 23 | 12 | 5 | 27 | 16 | 5 | 11 | 14
  Grade 3 Fatigue, Dose 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Related Fatigue, Dose 1 | 21 | 8 | 4 | 24 | 14 | 5 | 7 | 11
  Any Headache, Dose 1 | 20 | 11 | 5 | 14 | 18 | 5 | 6 | 11
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Headache, Dose 1 | 17 | 7 | 4 | 12 | 12 | 3 | 6 | 10
  Any Joint pain at other location, Dose 1 | 11 | 7 | 4 | 11 | 7 | 3 | 1 | 6
  Grade 3 Joint pain at other location, Dose 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Related Joint pain at other location, Dose 1 | 10 | 5 | 3 | 10 | 6 | 3 | 0 | 4
  Any Muscle aches, Dose 1 | 25 | 11 | 4 | 29 | 16 | 6 | 7 | 4
  Grade 3 Muscle aches, Dose 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Muscle aches, Dose 1 | 22 | 9 | 2 | 25 | 11 | 5 | 5 | 3
  Any Shivering, Dose 1 | 6 | 5 | 2 | 4 | 4 | 3 | 2 | 7
  Grade 3 Shivering, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Related Shivering, Dose 1 | 4 | 3 | 2 | 4 | 2 | 2 | 2 | 6
  Any Sweating, Dose 1 | 3 | 2 | 1 | 3 | 4 | 0 | 1 | 2
  Grade 3 Sweating, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating, Dose 1 | 3 | 1 | 0 | 3 | 4 | 0 | 1 | 2
  Any Temperature, Dose 1 | 1 | 0 | 0 | 2 | 4 | 2 | 2 | 0
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Related Temperature, Dose 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Fatigue, Dose 2 | 29 | 12 | 3 | 15 | 17 | 4 | 8 | 11
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Fatigue, Dose 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Related Fatigue, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Fatigue, Dose 2 | 28 | 12 | 1 | 10 | 11 | 3 | 6 | 8
  Any Headache, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Headache, Dose 2 | 23 | 7 | 5 | 12 | 10 | 1 | 7 | 12
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Headache, Dose 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Headache, Dose 2 | 20 | 7 | 2 | 9 | 4 | 1 | 7 | 7
  Any Joint pain at other location, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Joint pain at other location, Dose 2 | 16 | 12 | 2 | 12 | 9 | 2 | 3 | 5
  Grade 3 Joint pain at other location, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Joint pain at other location, Dose 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Related Joint pain at other location, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Joint pain at other location, Dose 2 | 15 | 12 | 2 | 9 | 4 | 2 | 2 | 4
  Any Muscle aches, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Muscle aches, Dose 2 | 30 | 17 | 2 | 11 | 13 | 4 | 5 | 8
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Muscle aches, Dose 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Muscle aches, Dose 2 | 27 | 17 | 1 | 8 | 8 | 4 | 3 | 7
  Any Shivering, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Shivering, Dose 2 | 8 | 5 | 0 | 2 | 6 | 3 | 1 | 6
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Shivering, Dose 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Shivering, Dose 2 | 7 | 5 | 0 | 1 | 5 | 3 | 1 | 5
  Any Sweating, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Sweating, Dose 2 | 6 | 2 | 1 | 1 | 3 | 2 | 0 | 1
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Sweating, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Sweating, Dose 2 | 5 | 2 | 0 | 0 | 3 | 1 | 0 | 1
  Any Temperature, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Any Temperature, Dose 2 | 1 | 0 | 1 | 2 | 4 | 1 | 0 | 2
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 126 | 66 | 63 | 130 | 129 | 65 | 63 | 130
  Related Temperature, Dose 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Any Fatigue, Across doses | 38 | 18 | 6 | 31 | 28 | 8 | 17 | 20
  Grade 3 Fatigue, Across doses | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 2
  Related Fatigue, Across doses | 36 | 15 | 4 | 27 | 21 | 7 | 11 | 15
  Any Headache, Across doses | 34 | 13 | 9 | 23 | 25 | 6 | 11 | 17
  Grade 3 Headache, Across doses | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Related Headache, Across doses | 29 | 10 | 6 | 19 | 15 | 4 | 11 | 13
  Any Joint pain at other location, Across doses | 22 | 14 | 5 | 18 | 15 | 4 | 3 | 9
  Grade 3 Joint pain at other location, Across doses | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Related Joint pain at other location, Across doses | 20 | 13 | 4 | 17 | 9 | 4 | 2 | 6
  Any Muscle aches, Across doses | 41 | 18 | 6 | 31 | 23 | 10 | 11 | 9
  Grade 3 Muscle aches, Across doses | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Related Muscle aches, Across doses | 35 | 18 | 3 | 27 | 17 | 9 | 8 | 7
  Any Shivering, Across doses | 13 | 9 | 2 | 5 | 10 | 6 | 2 | 13
  Grade 3 Shivering, Across doses | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Related Shivering, Across doses | 10 | 7 | 2 | 5 | 7 | 5 | 2 | 11
  Any Sweating, Across doses | 8 | 4 | 1 | 4 | 7 | 2 | 1 | 3
  Grade 3 Sweating, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Sweating, Across doses | 7 | 3 | 0 | 3 | 7 | 1 | 1 | 3
  Any Temperature, Across doses | 2 | 0 | 1 | 3 | 7 | 2 | 2 | 2
  Grade 3 Temperature, Across doses | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Related Temperature, Across doses | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1

38. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Results were tabulated for subjects in GSK2340273A F2_1D Group, who were older than 60 years of age (>60y).
Time Frame: During the 7-day (Days 0-6) post-Dose 3 vaccination period, for subjects > 60 years of age
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received at least 1 study vaccination and had their symptom sheets filled in. This analysis focused on subjects who received an additional dose of GSK2340273A F2 vaccine from GSK2340273A F2_1D Group.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340273A F2_1D Group
Number analyzed (Participants) | 64
Participants
  Any Pain | 6
  Grade 3 Pain | 0
  Any Redness | 1
  Grade 3 Redness | 0
  Any Swelling | 0
  Grade 3 Swelling | 0

39. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)], headache, joint pain at other location, muscle aches, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Results were tabulated for subjects in GSK2340273A F2_1D Group, who were older than 60 years of age (>60y).
Time Frame: During the 7-day (Days 0-6) post-Dose 3 vaccination period, for subjects > 60 years of age
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340273A F2_1D Group
Number analyzed (Participants) | 63
Participants
  Any Fatigue | 6
  Grade 3 Fatigue | 0
  Related Fatigue | 6
  Any Headache | 6
  Grade 3 Headache | 0
  Related Headache | 4
  Any Joint pain at other location | 3
  Grade 3 Joint pain at other location | 0
  Related Joint pain at other location | 2
  Any Muscle aches | 4
  Grade 3 Muscle aches | 0
  Related Muscle aches | 3
  Any Shivering | 1
  Grade 3 Shivering | 0
  Related Shivering | 0
  Any Sweating | 1
  Grade 3 Sweating | 0
  Related Sweating | 1
  Any Temperature | 0
  Grade 3 Temperature | 0
  Related Temperature | 0

40. Secondary Outcome: Number of Subjects With Abnormal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], alkaline phosphatase [AP], aspartate aminotransferase [AST], basophils [BAS], bilirubin [BIL], bilirubin conjugated/direct [BIL/CD] creatinine [CREA], eosinophils [EOS], hematocrit [HEM], haemoglobin [Hgb], lymphocytes [LYM], monocytes [MON], neutrophils [NEU], platelets [PLA], red blood cells [RBC], blood urea nitrogen [BUN] and white blood cells [WBC].
  Levels of haematological/biochemical parameters assessed in terms of normal laboratory values were - unknown, below, within and above the reference range defined for the specified time point and laboratory parameter.
Time Frame: At Days 7, 21, 28, 42 and 182, for subjects between 18-64 years of age
Population: The analysis was performed on the Total Vaccinated cohort included all subjects who received at least 1 study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 49 | 47 | 92
Participants
  ALT, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALT, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 7: Within | 92 | 46 | 47 | 90 | 89 | 49 | 46 | 91
  ALT, Day 7: Above | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1
  ALT, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  ALT, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 21: Within | 92 | 47 | 45 | 89 | 89 | 48 | 46 | 92
  ALT, Day 21: Above | 1 | 0 | 2 | 2 | 3 | 0 | 1 | 0
  ALT, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  ALT, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 28: Within | 91 | 47 | 46 | 87 | 90 | 47 | 45 | 88
  ALT, Day 28: Above | 1 | 0 | 1 | 4 | 1 | 0 | 2 | 3
  ALT, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  ALT, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 42: Within | 90 | 45 | 44 | 88 | 89 | 48 | 45 | 87
  ALT, Day 42: Above | 2 | 1 | 2 | 3 | 2 | 0 | 2 | 3
  ALT, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  ALT, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 182: Within | 87 | 47 | 46 | 86 | 86 | 46 | 46 | 89
  ALT, Day 182: Above | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2
  AP, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AP, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 7: Within | 92 | 46 | 47 | 90 | 91 | 47 | 44 | 90
  AP, Day 7: Above | 1 | 1 | 0 | 1 | 0 | 2 | 3 | 2
  AP, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  AP, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 21: Within | 92 | 46 | 47 | 90 | 91 | 47 | 46 | 89
  AP, Day 21: Above | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 3
  AP, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  AP, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 28: Within | 91 | 46 | 47 | 90 | 89 | 46 | 46 | 89
  AP, Day 28: Above | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 2
  AP, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  AP, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AP, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 42: Within | 90 | 45 | 46 | 90 | 91 | 46 | 46 | 90
  AP, Day 42: Above | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0
  AP, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  AP, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 182: Within | 86 | 47 | 46 | 87 | 88 | 45 | 46 | 87
  AP, Day 182: Above | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 4
  AST, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 7: Within | 93 | 47 | 47 | 90 | 90 | 49 | 47 | 91
  AST, Day 7: Above | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  AST, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  AST, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 21: Within | 92 | 47 | 46 | 89 | 90 | 48 | 46 | 92
  AST, Day 21: Above | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 0
  AST, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  AST, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 28: Within | 91 | 46 | 47 | 90 | 90 | 47 | 46 | 88
  AST, Day 28: Above | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 3
  AST, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  AST, Day 42: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  AST, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 42: Within | 92 | 45 | 46 | 90 | 89 | 47 | 46 | 88
  AST, Day 42: Above | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2
  AST, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  AST, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 182: Within | 87 | 46 | 46 | 86 | 86 | 46 | 46 | 89
  AST, Day 182: Above | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2
  BAS, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 7: Within | 92 | 47 | 47 | 91 | 92 | 49 | 47 | 92
  BAS, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  BAS, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  BAS, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 21: Within | 93 | 47 | 47 | 91 | 91 | 46 | 47 | 91
  BAS, Day 21: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  BAS, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  BAS, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 28: Within | 92 | 47 | 47 | 91 | 90 | 47 | 47 | 90
  BAS, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  BAS, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  BAS, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 42: Within | 92 | 45 | 44 | 90 | 90 | 47 | 46 | 91
  BAS, Day 42: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  BAS, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  BAS, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 182: Within | 87 | 47 | 45 | 88 | 87 | 47 | 46 | 90
  BAS, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BIL, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 7: Within | 93 | 46 | 47 | 90 | 91 | 49 | 46 | 90
  BIL, Day 7: Above | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2
  BIL, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  BIL, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 21: Within | 91 | 45 | 46 | 91 | 92 | 48 | 46 | 91
  BIL, Day 21: Above | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 1
  BIL, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  BIL, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 28: Within | 92 | 46 | 46 | 88 | 89 | 47 | 46 | 88
  BIL, Day 28: Above | 0 | 1 | 1 | 3 | 2 | 0 | 1 | 3
  BIL, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  BIL, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BIL, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 42: Within | 90 | 46 | 45 | 88 | 91 | 48 | 46 | 88
  BIL, Day 42: Above | 2 | 0 | 1 | 3 | 0 | 0 | 1 | 2
  BIL, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  BIL, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 182: Within | 87 | 46 | 45 | 88 | 88 | 47 | 45 | 90
  BIL, Day 182: Above | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  BIL/CD, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BIL/CD, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 7: Within | 93 | 47 | 47 | 91 | 91 | 49 | 47 | 92
  BIL/CD, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  BIL/CD, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 21: Within | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  BIL/CD, Day 21: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  BIL/CD, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 28: Within | 92 | 47 | 47 | 91 | 91 | 47 | 46 | 91
  BIL/CD, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BIL/CD, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  BIL/CD, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BIL/CD, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 42: Within | 92 | 45 | 46 | 91 | 91 | 48 | 47 | 90
  BIL/CD, Day 42: Above | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  BIL/CD, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 182: Within | 87 | 47 | 46 | 88 | 88 | 47 | 45 | 90
  BIL/CD, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  CREA, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CREA, Day 7: Below | 5 | 1 | 4 | 2 | 8 | 2 | 3 | 6
  CREA, Day 7: Within | 88 | 45 | 43 | 86 | 83 | 47 | 44 | 85
  CREA, Day 7: Above | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1
  CREA, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  CREA, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Day 21: Below | 10 | 3 | 5 | 8 | 8 | 3 | 3 | 11
  CREA, Day 21: Within | 82 | 43 | 41 | 83 | 83 | 45 | 44 | 79
  CREA, Day 21: Above | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  CREA, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  CREA, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Day 28: Below | 9 | 1 | 4 | 4 | 12 | 4 | 3 | 9
  CREA, Day 28: Within | 82 | 46 | 42 | 87 | 77 | 42 | 44 | 82
  CREA, Day 28: Above | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
  CREA, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  CREA, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  CREA, Day 42: Below | 11 | 3 | 6 | 8 | 14 | 2 | 4 | 12
  CREA, Day 42: Within | 79 | 43 | 40 | 83 | 77 | 46 | 43 | 76
  CREA, Day 42: Above | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  CREA, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  CREA, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Day 182: Below | 7 | 2 | 9 | 7 | 13 | 3 | 6 | 10
  CREA, Day 182: Within | 79 | 44 | 37 | 81 | 75 | 44 | 40 | 79
  CREA, Day 182: Above | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  EOS, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Day 7: Below | 2 | 0 | 1 | 5 | 5 | 1 | 1 | 2
  EOS, Day 7: Within | 88 | 45 | 44 | 84 | 82 | 47 | 46 | 88
  EOS, Day 7: Above | 2 | 2 | 2 | 2 | 5 | 1 | 0 | 2
  EOS, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  EOS, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  EOS, Day 21: Below | 2 | 3 | 0 | 5 | 7 | 1 | 1 | 5
  EOS, Day 21: Within | 89 | 44 | 46 | 86 | 83 | 45 | 45 | 83
  EOS, Day 21: Above | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  EOS, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  EOS, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  EOS, Day 28: Below | 3 | 0 | 2 | 4 | 7 | 3 | 3 | 3
  EOS, Day 28: Within | 86 | 47 | 44 | 85 | 80 | 43 | 42 | 84
  EOS, Day 28: Above | 3 | 0 | 1 | 2 | 3 | 1 | 2 | 3
  EOS, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  EOS, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  EOS, Day 42: Below | 4 | 6 | 2 | 6 | 5 | 3 | 2 | 2
  EOS, Day 42: Within | 87 | 39 | 42 | 84 | 81 | 43 | 42 | 87
  EOS, Day 42: Above | 1 | 0 | 0 | 0 | 4 | 1 | 2 | 2
  EOS, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  EOS, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  EOS, Day 182: Below | 1 | 4 | 4 | 2 | 4 | 2 | 3 | 3
  EOS, Day 182: Within | 85 | 42 | 41 | 86 | 80 | 43 | 41 | 86
  EOS, Day 182: Above | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 1
  HEM, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEM, Day 7: Below | 1 | 2 | 0 | 3 | 3 | 0 | 0 | 2
  HEM, Day 7: Within | 89 | 43 | 46 | 85 | 89 | 48 | 47 | 88
  HEM, Day 7: Above | 2 | 2 | 1 | 3 | 0 | 1 | 0 | 2
  HEM, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  HEM, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  HEM, Day 21: Below | 2 | 1 | 1 | 3 | 4 | 3 | 1 | 3
  HEM, Day 21: Within | 88 | 43 | 46 | 85 | 88 | 43 | 45 | 89
  HEM, Day 21: Above | 3 | 3 | 0 | 3 | 0 | 0 | 1 | 0
  HEM, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  HEM, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEM, Day 28: Below | 5 | 4 | 1 | 3 | 2 | 1 | 2 | 4
  HEM, Day 28: Within | 85 | 42 | 45 | 86 | 88 | 46 | 45 | 85
  HEM, Day 28: Above | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 2
  HEM, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  HEM, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  HEM, Day 42: Below | 8 | 1 | 2 | 4 | 7 | 1 | 3 | 3
  HEM, Day 42: Within | 83 | 44 | 41 | 83 | 83 | 46 | 43 | 88
  HEM, Day 42: Above | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
  HEM, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  HEM, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  HEM, Day 182: Below | 2 | 3 | 0 | 6 | 7 | 2 | 4 | 6
  HEM, Day 182: Within | 85 | 44 | 44 | 81 | 79 | 45 | 41 | 83
  HEM, Day 182: Above | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
  HgB, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HgB, Day 7: Below | 3 | 0 | 2 | 5 | 5 | 1 | 0 | 3
  HgB, Day 7: Within | 89 | 46 | 44 | 84 | 87 | 48 | 47 | 88
  HgB, Day 7: Above | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1
  HgB, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  HgB, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  HgB, Day 21: Below | 5 | 1 | 0 | 5 | 6 | 2 | 2 | 1
  HgB, Day 21: Within | 88 | 45 | 47 | 84 | 86 | 44 | 44 | 91
  HgB, Day 21: Above | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
  HgB, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  HgB, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HgB, Day 28: Below | 7 | 3 | 1 | 2 | 2 | 1 | 2 | 4
  HgB, Day 28: Within | 85 | 44 | 45 | 88 | 88 | 46 | 45 | 85
  HgB, Day 28: Above | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  HgB, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  HgB, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  HgB, Day 42: Below | 6 | 2 | 1 | 3 | 3 | 0 | 2 | 4
  HgB, Day 42: Within | 85 | 42 | 42 | 84 | 86 | 47 | 43 | 86
  HgB, Day 42: Above | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 1
  HgB, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  HgB, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  HgB, Day 182: Below | 3 | 3 | 0 | 6 | 3 | 2 | 4 | 3
  HgB, Day 182: Within | 83 | 44 | 44 | 81 | 83 | 44 | 42 | 86
  HgB, Day 182: Above | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1
  LYM, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  LYM, Day 7: Within | 91 | 46 | 47 | 90 | 92 | 49 | 46 | 90
  LYM, Day 7: Above | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  LYM, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  LYM, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  LYM, Day 21: Below | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  LYM, Day 21: Within | 92 | 47 | 47 | 89 | 90 | 46 | 46 | 90
  LYM, Day 21: Above | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  LYM, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  LYM, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  LYM, Day 28: Below | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  LYM, Day 28: Within | 90 | 46 | 47 | 89 | 89 | 47 | 46 | 87
  LYM, Day 28: Above | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 3
  LYM, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  LYM, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  LYM, Day 42: Below | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  LYM, Day 42: Within | 89 | 45 | 42 | 89 | 89 | 47 | 45 | 90
  LYM, Day 42: Above | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  LYM, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  LYM, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  LYM, Day 182: Below | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  LYM, Day 182: Within | 86 | 47 | 45 | 87 | 86 | 46 | 43 | 88
  LYM, Day 182: Above | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
  MON, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MON, Day 7: Below | 21 | 11 | 10 | 17 | 16 | 8 | 4 | 13
  MON, Day 7: Within | 71 | 36 | 37 | 74 | 76 | 41 | 43 | 78
  MON, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MON, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  MON, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  MON, Day 21: Below | 21 | 14 | 8 | 18 | 21 | 6 | 8 | 23
  MON, Day 21: Within | 72 | 33 | 39 | 73 | 70 | 40 | 39 | 68
  MON, Day 21: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MON, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  MON, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  MON, Day 28: Below | 27 | 11 | 6 | 21 | 12 | 8 | 9 | 18
  MON, Day 28: Within | 65 | 36 | 41 | 70 | 78 | 39 | 38 | 72
  MON, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MON, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  MON, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  MON, Day 42: Below | 29 | 8 | 9 | 17 | 15 | 9 | 7 | 15
  MON, Day 42: Within | 62 | 37 | 35 | 73 | 75 | 38 | 39 | 76
  MON, Day 42: Above | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MON, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  MON, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  MON, Day 182: Below | 18 | 11 | 8 | 18 | 19 | 13 | 7 | 19
  MON, Day 182: Within | 69 | 36 | 37 | 70 | 68 | 34 | 39 | 71
  MON, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Day 7: Below | 3 | 2 | 1 | 1 | 0 | 1 | 2 | 1
  NEU, Day 7: Within | 87 | 45 | 45 | 87 | 91 | 47 | 44 | 89
  NEU, Day 7: Above | 2 | 0 | 1 | 3 | 1 | 1 | 1 | 2
  NEU, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  NEU, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  NEU, Day 21: Below | 5 | 1 | 2 | 2 | 1 | 1 | 0 | 4
  NEU, Day 21: Within | 86 | 45 | 45 | 88 | 89 | 45 | 46 | 85
  NEU, Day 21: Above | 2 | 1 | 0 | 1 | 1 | 0 | 1 | 2
  NEU, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  NEU, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  NEU, Day 28: Below | 4 | 5 | 1 | 4 | 1 | 0 | 2 | 2
  NEU, Day 28: Within | 84 | 41 | 45 | 87 | 88 | 47 | 45 | 88
  NEU, Day 28: Above | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  NEU, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  NEU, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  NEU, Day 42: Below | 7 | 5 | 1 | 1 | 0 | 1 | 2 | 2
  NEU, Day 42: Within | 82 | 40 | 43 | 88 | 89 | 46 | 42 | 87
  NEU, Day 42: Above | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 2
  NEU, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  NEU, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  NEU, Day 182: Below | 4 | 5 | 2 | 2 | 1 | 1 | 2 | 4
  NEU, Day 182: Within | 82 | 41 | 43 | 86 | 85 | 46 | 41 | 85
  NEU, Day 182: Above | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1
  PLA, Day 7: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  PLA, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Day 7: Within | 91 | 47 | 47 | 91 | 91 | 49 | 46 | 90
  PLA, Day 7: Above | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  PLA, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  PLA, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  PLA, Day 21: Below | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Day 21: Within | 91 | 47 | 47 | 90 | 92 | 46 | 46 | 92
  PLA, Day 21: Above | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  PLA, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  PLA, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  PLA, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Day 28: Within | 91 | 47 | 47 | 91 | 89 | 47 | 46 | 91
  PLA, Day 28: Above | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLA, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  PLA, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  PLA, Day 42: Below | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  PLA, Day 42: Within | 91 | 44 | 44 | 90 | 89 | 47 | 46 | 91
  PLA, Day 42: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  PLA, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  PLA, Day 182: Below | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Day 182: Within | 86 | 47 | 44 | 87 | 87 | 46 | 46 | 90
  PLA, Day 182: Above | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  RBC, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Day 7: Below | 1 | 2 | 1 | 3 | 5 | 2 | 4 | 3
  RBC, Day 7: Within | 90 | 44 | 46 | 86 | 86 | 47 | 43 | 89
  RBC, Day 7: Above | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0
  RBC, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  RBC, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  RBC, Day 21: Below | 4 | 1 | 2 | 3 | 3 | 2 | 5 | 6
  RBC, Day 21: Within | 88 | 45 | 45 | 88 | 87 | 43 | 42 | 86
  RBC, Day 21: Above | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
  RBC, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  RBC, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  RBC, Day 28: Below | 3 | 4 | 3 | 3 | 3 | 1 | 3 | 7
  RBC, Day 28: Within | 88 | 42 | 44 | 87 | 86 | 46 | 44 | 84
  RBC, Day 28: Above | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  RBC, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  RBC, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  RBC, Day 42: Below | 6 | 3 | 4 | 2 | 5 | 0 | 3 | 5
  RBC, Day 42: Within | 85 | 41 | 40 | 87 | 85 | 47 | 43 | 86
  RBC, Day 42: Above | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  RBC, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  RBC, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  RBC, Day 182: Below | 7 | 3 | 2 | 10 | 3 | 1 | 4 | 9
  RBC, Day 182: Within | 79 | 44 | 43 | 78 | 82 | 46 | 42 | 81
  RBC, Day 182: Above | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  BUN, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, Day 7: Below | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  BUN, Day 7: Within | 92 | 47 | 46 | 91 | 89 | 48 | 47 | 90
  BUN, Day 7: Above | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  BUN, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  BUN, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 21: Below | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  BUN, Day 21: Within | 91 | 46 | 46 | 89 | 90 | 47 | 45 | 89
  BUN, Day 21: Above | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 2
  BUN, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  BUN, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 28: Below | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  BUN, Day 28: Within | 89 | 47 | 46 | 89 | 89 | 46 | 47 | 91
  BUN, Day 28: Above | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  BUN, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  BUN, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BUN, Day 42: Below | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  BUN, Day 42: Within | 90 | 46 | 45 | 89 | 91 | 48 | 46 | 90
  BUN, Day 42: Above | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  BUN, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  BUN, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 182: Below | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  BUN, Day 182: Within | 85 | 44 | 44 | 88 | 87 | 46 | 46 | 91
  BUN, Day 182: Above | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
  WBC, Day 7: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Day 7: Below | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 2
  WBC, Day 7: Within | 88 | 45 | 45 | 86 | 90 | 48 | 44 | 87
  WBC, Day 7: Above | 1 | 0 | 1 | 5 | 1 | 1 | 2 | 3
  WBC, Day 21: number analyzed (Participants) | 93 | 47 | 47 | 91 | 92 | 48 | 47 | 92
  WBC, Day 21: Unknown | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  WBC, Day 21: Below | 5 | 1 | 2 | 2 | 2 | 0 | 0 | 4
  WBC, Day 21: Within | 86 | 45 | 45 | 86 | 87 | 46 | 46 | 84
  WBC, Day 21: Above | 2 | 1 | 0 | 3 | 2 | 0 | 1 | 3
  WBC, Day 28: number analyzed (Participants) | 92 | 47 | 47 | 91 | 91 | 47 | 47 | 91
  WBC, Day 28: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  WBC, Day 28: Below | 5 | 4 | 1 | 3 | 1 | 1 | 1 | 2
  WBC, Day 28: Within | 84 | 42 | 44 | 87 | 88 | 46 | 44 | 86
  WBC, Day 28: Above | 3 | 1 | 2 | 1 | 1 | 0 | 2 | 2
  WBC, Day 42: number analyzed (Participants) | 92 | 46 | 46 | 91 | 91 | 48 | 47 | 91
  WBC, Day 42: Unknown | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  WBC, Day 42: Below | 6 | 4 | 0 | 2 | 2 | 2 | 1 | 4
  WBC, Day 42: Within | 82 | 41 | 43 | 87 | 87 | 45 | 44 | 85
  WBC, Day 42: Above | 4 | 0 | 1 | 1 | 1 | 0 | 1 | 2
  WBC, Day 182: number analyzed (Participants) | 88 | 47 | 46 | 88 | 88 | 47 | 46 | 91
  WBC, Day 182: Unknown | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  WBC, Day 182: Below | 7 | 4 | 2 | 2 | 2 | 0 | 1 | 6
  WBC, Day 182: Within | 79 | 42 | 42 | 85 | 84 | 46 | 42 | 81
  WBC, Day 182: Above | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3

41. Secondary Outcome: Number of Subjects With Abnormal Biochemical and Haematological Levels
Description: as for outcome 40
Time Frame: At Days 7, 21, 28, 42 and 182, for subjects > 64 years of age
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received at least 1 study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 64 | 130
Participants
  ALT, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  ALT, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ALT, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 7: Within | 126 | 66 | 65 | 127 | 129 | 65 | 63 | 130
  ALT, Day 7: Above | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  ALT, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  ALT, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALT, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 21: Within | 126 | 66 | 62 | 128 | 128 | 64 | 63 | 128
  ALT, Day 21: Above | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 1
  ALT, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  ALT, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  ALT, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 28: Within | 126 | 65 | 63 | 126 | 125 | 64 | 60 | 127
  ALT, Day 28: Above | 1 | 0 | 0 | 3 | 4 | 1 | 2 | 2
  ALT, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  ALT, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 42: Within | 128 | 65 | 62 | 127 | 125 | 65 | 63 | 128
  ALT, Day 42: Above | 0 | 0 | 1 | 3 | 4 | 0 | 0 | 2
  ALT, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  ALT, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALT, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Day 182: Within | 123 | 63 | 63 | 128 | 126 | 65 | 63 | 130
  ALT, Day 182: Above | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  AP, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  AP, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AP, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 7: Within | 126 | 66 | 64 | 127 | 127 | 64 | 62 | 129
  AP, Day 7: Above | 2 | 0 | 1 | 2 | 3 | 1 | 1 | 1
  AP, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  AP, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AP, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 21: Within | 125 | 66 | 61 | 130 | 128 | 62 | 63 | 127
  AP, Day 21: Above | 2 | 0 | 2 | 0 | 2 | 2 | 1 | 2
  AP, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  AP, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  AP, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 28: Within | 121 | 65 | 61 | 129 | 128 | 64 | 61 | 125
  AP, Day 28: Above | 6 | 0 | 2 | 0 | 1 | 1 | 1 | 4
  AP, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  AP, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 42: Within | 122 | 65 | 61 | 129 | 125 | 64 | 62 | 128
  AP, Day 42: Above | 6 | 0 | 2 | 1 | 4 | 1 | 1 | 2
  AP, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  AP, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AP, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AP, Day 182: Within | 123 | 63 | 62 | 128 | 125 | 64 | 63 | 130
  AP, Day 182: Above | 2 | 0 | 1 | 1 | 3 | 1 | 0 | 0
  AST, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  AST, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  AST, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 7: Within | 128 | 66 | 65 | 128 | 129 | 65 | 63 | 130
  AST, Day 7: Above | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  AST, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  AST, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AST, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 21: Within | 127 | 66 | 62 | 130 | 129 | 64 | 64 | 128
  AST, Day 21: Above | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  AST, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  AST, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  AST, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 28: Within | 127 | 65 | 63 | 128 | 129 | 65 | 61 | 129
  AST, Day 28: Above | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  AST, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  AST, Day 42: Unknown | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  AST, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 42: Within | 128 | 65 | 62 | 128 | 127 | 65 | 63 | 130
  AST, Day 42: Above | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  AST, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  AST, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  AST, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Day 182: Within | 124 | 63 | 63 | 129 | 126 | 64 | 63 | 130
  AST, Day 182: Above | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  BAS, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  BAS, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  BAS, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 7: Within | 129 | 66 | 65 | 129 | 127 | 65 | 63 | 130
  BAS, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  BAS, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  BAS, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 21: Within | 126 | 66 | 63 | 129 | 128 | 65 | 62 | 129
  BAS, Day 21: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  BAS, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  BAS, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 28: Within | 127 | 66 | 63 | 130 | 129 | 65 | 63 | 128
  BAS, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  BAS, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  BAS, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 42: Within | 125 | 63 | 61 | 130 | 127 | 64 | 63 | 128
  BAS, Day 42: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  BAS, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  BAS, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Day 182: Within | 125 | 63 | 62 | 129 | 129 | 65 | 63 | 130
  BAS, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  BIL, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  BIL, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 7: Within | 126 | 66 | 65 | 128 | 130 | 65 | 63 | 129
  BIL, Day 7: Above | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  BIL, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  BIL, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BIL, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 21: Within | 126 | 66 | 62 | 129 | 130 | 64 | 64 | 129
  BIL, Day 21: Above | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  BIL, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  BIL, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  BIL, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 28: Within | 126 | 65 | 63 | 128 | 129 | 65 | 62 | 127
  BIL, Day 28: Above | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  BIL, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  BIL, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 42: Within | 126 | 65 | 63 | 129 | 127 | 65 | 63 | 128
  BIL, Day 42: Above | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2
  BIL, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  BIL, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BIL, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL, Day 182: Within | 124 | 63 | 63 | 129 | 127 | 65 | 63 | 129
  BIL, Day 182: Above | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  BIL/CD, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  BIL/CD, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  BIL/CD, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 7: Within | 128 | 66 | 65 | 129 | 130 | 65 | 63 | 130
  BIL/CD, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  BIL/CD, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BIL/CD, Day 21: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 21: Within | 127 | 66 | 63 | 130 | 130 | 64 | 64 | 129
  BIL/CD, Day 21: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  BIL/CD, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  BIL/CD, Day 28: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 28: Within | 127 | 65 | 63 | 129 | 129 | 65 | 62 | 129
  BIL/CD, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  BIL/CD, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 42: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 42: Within | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  BIL/CD, Day 42: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  BIL/CD, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BIL/CD, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BIL/CD, Day 182: Within | 125 | 63 | 63 | 129 | 128 | 65 | 63 | 130
  BIL/CD, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  CREA, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  CREA, Day 7: Below | 6 | 7 | 5 | 11 | 10 | 4 | 5 | 5
  CREA, Day 7: Within | 119 | 59 | 60 | 117 | 120 | 61 | 57 | 124
  CREA, Day 7: Above | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  CREA, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  CREA, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  CREA, Day 21: Below | 13 | 7 | 7 | 12 | 7 | 6 | 4 | 6
  CREA, Day 21: Within | 112 | 59 | 56 | 118 | 122 | 57 | 59 | 119
  CREA, Day 21: Above | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 4
  CREA, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  CREA, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  CREA, Day 28: Below | 8 | 6 | 7 | 14 | 7 | 6 | 5 | 6
  CREA, Day 28: Within | 118 | 59 | 56 | 113 | 122 | 58 | 56 | 121
  CREA, Day 28: Above | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 2
  CREA, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  CREA, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Day 42: Below | 12 | 5 | 7 | 12 | 8 | 5 | 6 | 9
  CREA, Day 42: Within | 115 | 60 | 54 | 118 | 121 | 58 | 56 | 119
  CREA, Day 42: Above | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 2
  CREA, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  CREA, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  CREA, Day 182: Below | 15 | 7 | 5 | 15 | 7 | 5 | 5 | 11
  CREA, Day 182: Within | 107 | 56 | 58 | 110 | 120 | 60 | 56 | 119
  CREA, Day 182: Above | 3 | 0 | 0 | 4 | 1 | 0 | 2 | 0
  EOS, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  EOS, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  EOS, Day 7: Below | 4 | 1 | 1 | 4 | 1 | 3 | 3 | 5
  EOS, Day 7: Within | 123 | 64 | 61 | 121 | 120 | 61 | 56 | 122
  EOS, Day 7: Above | 2 | 1 | 3 | 4 | 6 | 1 | 4 | 3
  EOS, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  EOS, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  EOS, Day 21: Below | 3 | 0 | 0 | 3 | 5 | 1 | 4 | 5
  EOS, Day 21: Within | 119 | 65 | 60 | 121 | 116 | 62 | 56 | 119
  EOS, Day 21: Above | 4 | 1 | 3 | 5 | 7 | 2 | 2 | 5
  EOS, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  EOS, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  EOS, Day 28: Below | 2 | 0 | 1 | 5 | 5 | 4 | 4 | 6
  EOS, Day 28: Within | 122 | 63 | 58 | 120 | 120 | 57 | 56 | 118
  EOS, Day 28: Above | 3 | 3 | 4 | 5 | 4 | 4 | 3 | 4
  EOS, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  EOS, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  EOS, Day 42: Below | 4 | 0 | 1 | 1 | 2 | 2 | 6 | 8
  EOS, Day 42: Within | 116 | 62 | 57 | 123 | 123 | 60 | 55 | 116
  EOS, Day 42: Above | 5 | 1 | 3 | 6 | 2 | 2 | 2 | 4
  EOS, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  EOS, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  EOS, Day 182: Below | 7 | 0 | 2 | 7 | 2 | 0 | 3 | 6
  EOS, Day 182: Within | 112 | 62 | 56 | 117 | 124 | 62 | 58 | 119
  EOS, Day 182: Above | 6 | 1 | 4 | 5 | 3 | 3 | 2 | 5
  HEM, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  HEM, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HEM, Day 7: Below | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
  HEM, Day 7: Within | 127 | 66 | 65 | 126 | 125 | 64 | 60 | 124
  HEM, Day 7: Above | 2 | 0 | 0 | 2 | 3 | 1 | 2 | 6
  HEM, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  HEM, Day 21: Unknown | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  HEM, Day 21: Below | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 2
  HEM, Day 21: Within | 125 | 63 | 62 | 126 | 121 | 64 | 61 | 121
  HEM, Day 21: Above | 2 | 3 | 0 | 2 | 4 | 0 | 2 | 6
  HEM, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  HEM, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HEM, Day 28: Below | 1 | 0 | 1 | 1 | 4 | 1 | 1 | 1
  HEM, Day 28: Within | 123 | 65 | 62 | 127 | 122 | 64 | 61 | 123
  HEM, Day 28: Above | 3 | 1 | 0 | 2 | 3 | 0 | 1 | 5
  HEM, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  HEM, Day 42: Unknown | 3 | 2 | 1 | 0 | 2 | 1 | 0 | 2
  HEM, Day 42: Below | 2 | 0 | 0 | 2 | 4 | 1 | 2 | 3
  HEM, Day 42: Within | 120 | 63 | 62 | 127 | 118 | 63 | 60 | 121
  HEM, Day 42: Above | 3 | 0 | 0 | 1 | 5 | 0 | 1 | 4
  HEM, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  HEM, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEM, Day 182: Below | 5 | 0 | 2 | 0 | 2 | 0 | 1 | 8
  HEM, Day 182: Within | 118 | 62 | 60 | 128 | 126 | 65 | 61 | 118
  HEM, Day 182: Above | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 4
  HgB, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  HgB, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HgB, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HgB, Day 7: Within | 127 | 66 | 65 | 128 | 129 | 65 | 60 | 128
  HgB, Day 7: Above | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2
  HgB, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  HgB, Day 21: Unknown | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  HgB, Day 21: Below | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 2
  HgB, Day 21: Within | 122 | 66 | 63 | 127 | 124 | 65 | 59 | 123
  HgB, Day 21: Above | 3 | 0 | 0 | 3 | 2 | 0 | 2 | 4
  HgB, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  HgB, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HgB, Day 28: Below | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  HgB, Day 28: Within | 122 | 66 | 63 | 128 | 127 | 64 | 61 | 126
  HgB, Day 28: Above | 4 | 0 | 0 | 2 | 1 | 0 | 1 | 3
  HgB, Day 42: number analyzed (Participants) | 128 | 65 | 62 | 130 | 129 | 65 | 63 | 130
  HgB, Day 42: Unknown | 3 | 2 | 0 | 0 | 2 | 1 | 0 | 2
  HgB, Day 42: Below | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3
  HgB, Day 42: Within | 121 | 63 | 61 | 128 | 122 | 63 | 60 | 122
  HgB, Day 42: Above | 3 | 0 | 1 | 2 | 4 | 0 | 1 | 3
  HgB, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  HgB, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HgB, Day 182: Below | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 5
  HgB, Day 182: Within | 123 | 63 | 59 | 128 | 126 | 65 | 61 | 120
  HgB, Day 182: Above | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 5
  LYM, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  LYM, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  LYM, Day 7: Below | 3 | 1 | 0 | 0 | 2 | 2 | 1 | 3
  LYM, Day 7: Within | 126 | 65 | 65 | 129 | 124 | 63 | 61 | 126
  LYM, Day 7: Above | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  LYM, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  LYM, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  LYM, Day 21: Below | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 2
  LYM, Day 21: Within | 123 | 64 | 63 | 128 | 126 | 64 | 60 | 127
  LYM, Day 21: Above | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LYM, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  LYM, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  LYM, Day 28: Below | 4 | 2 | 0 | 2 | 0 | 3 | 0 | 3
  LYM, Day 28: Within | 121 | 64 | 63 | 127 | 129 | 62 | 63 | 124
  LYM, Day 28: Above | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  LYM, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  LYM, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  LYM, Day 42: Below | 4 | 3 | 1 | 1 | 5 | 2 | 1 | 3
  LYM, Day 42: Within | 120 | 59 | 60 | 128 | 120 | 61 | 62 | 125
  LYM, Day 42: Above | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0
  LYM, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  LYM, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYM, Day 182: Below | 4 | 1 | 1 | 0 | 0 | 2 | 0 | 1
  LYM, Day 182: Within | 121 | 61 | 61 | 128 | 127 | 63 | 63 | 129
  LYM, Day 182: Above | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
  MON, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  MON, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  MON, Day 7: Below | 20 | 6 | 12 | 12 | 13 | 3 | 9 | 15
  MON, Day 7: Within | 109 | 60 | 53 | 117 | 114 | 62 | 54 | 115
  MON, Day 7: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MON, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  MON, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  MON, Day 21: Below | 11 | 10 | 9 | 20 | 16 | 11 | 8 | 14
  MON, Day 21: Within | 115 | 56 | 54 | 108 | 112 | 54 | 54 | 115
  MON, Day 21: Above | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  MON, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  MON, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  MON, Day 28: Below | 15 | 10 | 6 | 15 | 15 | 8 | 3 | 19
  MON, Day 28: Within | 112 | 56 | 57 | 115 | 114 | 57 | 60 | 108
  MON, Day 28: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MON, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  MON, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  MON, Day 42: Below | 13 | 4 | 8 | 13 | 12 | 5 | 5 | 20
  MON, Day 42: Within | 112 | 59 | 53 | 117 | 114 | 59 | 58 | 108
  MON, Day 42: Above | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  MON, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  MON, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  MON, Day 182: Below | 14 | 7 | 7 | 21 | 15 | 9 | 7 | 21
  MON, Day 182: Within | 111 | 56 | 55 | 108 | 114 | 56 | 56 | 109
  MON, Day 182: Above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  NEU, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  NEU, Day 7: Below | 3 | 0 | 2 | 3 | 2 | 1 | 1 | 1
  NEU, Day 7: Within | 125 | 65 | 62 | 125 | 124 | 63 | 62 | 129
  NEU, Day 7: Above | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
  NEU, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  NEU, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  NEU, Day 21: Below | 4 | 2 | 1 | 2 | 5 | 3 | 3 | 1
  NEU, Day 21: Within | 119 | 63 | 62 | 124 | 122 | 62 | 58 | 126
  NEU, Day 21: Above | 3 | 1 | 0 | 3 | 1 | 0 | 1 | 2
  NEU, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  NEU, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  NEU, Day 28: Below | 3 | 1 | 0 | 3 | 2 | 1 | 2 | 0
  NEU, Day 28: Within | 121 | 65 | 62 | 124 | 126 | 62 | 61 | 125
  NEU, Day 28: Above | 3 | 0 | 1 | 3 | 1 | 2 | 0 | 3
  NEU, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  NEU, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  NEU, Day 42: Below | 3 | 1 | 1 | 3 | 4 | 1 | 1 | 3
  NEU, Day 42: Within | 119 | 62 | 60 | 126 | 123 | 63 | 61 | 123
  NEU, Day 42: Above | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  NEU, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  NEU, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  NEU, Day 182: Below | 4 | 0 | 2 | 3 | 4 | 2 | 1 | 0
  NEU, Day 182: Within | 120 | 62 | 58 | 124 | 125 | 62 | 61 | 130
  NEU, Day 182: Above | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 0
  PLA, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  PLA, Day 7: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  PLA, Day 7: Below | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 3
  PLA, Day 7: Within | 127 | 66 | 64 | 127 | 129 | 63 | 63 | 123
  PLA, Day 7: Above | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  PLA, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  PLA, Day 21: Unknown | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1
  PLA, Day 21: Below | 2 | 0 | 0 | 2 | 1 | 2 | 0 | 1
  PLA, Day 21: Within | 124 | 66 | 63 | 126 | 127 | 63 | 62 | 124
  PLA, Day 21: Above | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
  PLA, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  PLA, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  PLA, Day 28: Below | 2 | 0 | 1 | 2 | 3 | 0 | 0 | 1
  PLA, Day 28: Within | 125 | 66 | 62 | 125 | 126 | 65 | 62 | 124
  PLA, Day 28: Above | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2
  PLA, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  PLA, Day 42: Unknown | 3 | 2 | 1 | 0 | 2 | 1 | 0 | 3
  PLA, Day 42: Below | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 2
  PLA, Day 42: Within | 124 | 63 | 61 | 126 | 126 | 63 | 62 | 122
  PLA, Day 42: Above | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  PLA, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  PLA, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  PLA, Day 182: Below | 3 | 1 | 2 | 3 | 2 | 2 | 1 | 2
  PLA, Day 182: Within | 122 | 61 | 61 | 125 | 126 | 63 | 62 | 124
  PLA, Day 182: Above | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3
  RBC, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  RBC, Day 7: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  RBC, Day 7: Below | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0
  RBC, Day 7: Within | 127 | 64 | 64 | 130 | 125 | 64 | 60 | 129
  RBC, Day 7: Above | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 1
  RBC, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  RBC, Day 21: Unknown | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  RBC, Day 21: Below | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 1
  RBC, Day 21: Within | 124 | 64 | 63 | 129 | 124 | 65 | 60 | 127
  RBC, Day 21: Above | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 1
  RBC, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  RBC, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  RBC, Day 28: Below | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 1
  RBC, Day 28: Within | 123 | 65 | 62 | 130 | 127 | 63 | 62 | 127
  RBC, Day 28: Above | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 1
  RBC, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  RBC, Day 42: Unknown | 3 | 2 | 1 | 0 | 2 | 1 | 0 | 2
  RBC, Day 42: Below | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 3
  RBC, Day 42: Within | 122 | 61 | 62 | 129 | 121 | 62 | 62 | 122
  RBC, Day 42: Above | 2 | 2 | 0 | 0 | 4 | 0 | 0 | 3
  RBC, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  RBC, Day 182: Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Day 182: Below | 3 | 0 | 0 | 1 | 0 | 1 | 2 | 3
  RBC, Day 182: Within | 120 | 62 | 63 | 128 | 127 | 64 | 61 | 124
  RBC, Day 182: Above | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 3
  BUN, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  BUN, Day 7: Unknown | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  BUN, Day 7: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 7: Within | 124 | 66 | 65 | 126 | 128 | 65 | 63 | 129
  BUN, Day 7: Above | 4 | 0 | 0 | 3 | 2 | 0 | 0 | 1
  BUN, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  BUN, Day 21: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BUN, Day 21: Below | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  BUN, Day 21: Within | 123 | 65 | 62 | 127 | 128 | 63 | 64 | 124
  BUN, Day 21: Above | 4 | 0 | 0 | 3 | 2 | 1 | 0 | 5
  BUN, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  BUN, Day 28: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
  BUN, Day 28: Below | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 28: Within | 124 | 63 | 63 | 127 | 126 | 64 | 62 | 128
  BUN, Day 28: Above | 3 | 1 | 0 | 2 | 3 | 1 | 0 | 1
  BUN, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  BUN, Day 42: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 42: Below | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BUN, Day 42: Within | 125 | 64 | 62 | 128 | 125 | 63 | 63 | 127
  BUN, Day 42: Above | 3 | 0 | 1 | 2 | 4 | 2 | 0 | 3
  BUN, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  BUN, Day 182: Unknown | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  BUN, Day 182: Below | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BUN, Day 182: Within | 121 | 63 | 60 | 124 | 125 | 65 | 63 | 128
  BUN, Day 182: Above | 4 | 0 | 3 | 5 | 3 | 0 | 0 | 1
  WBC, Day 7: number analyzed (Participants) | 129 | 66 | 65 | 130 | 130 | 65 | 63 | 130
  WBC, Day 7: Unknown | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
  WBC, Day 7: Below | 3 | 0 | 1 | 2 | 3 | 1 | 1 | 0
  WBC, Day 7: Within | 125 | 66 | 63 | 125 | 123 | 62 | 62 | 129
  WBC, Day 7: Above | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 1
  WBC, Day 21: number analyzed (Participants) | 127 | 66 | 63 | 130 | 130 | 65 | 64 | 129
  WBC, Day 21: Unknown | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  WBC, Day 21: Below | 6 | 2 | 1 | 3 | 5 | 3 | 2 | 2
  WBC, Day 21: Within | 116 | 63 | 62 | 122 | 123 | 62 | 59 | 125
  WBC, Day 21: Above | 4 | 1 | 0 | 4 | 0 | 0 | 1 | 2
  WBC, Day 28: number analyzed (Participants) | 127 | 66 | 63 | 130 | 129 | 65 | 64 | 129
  WBC, Day 28: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  WBC, Day 28: Below | 6 | 1 | 0 | 1 | 2 | 1 | 2 | 2
  WBC, Day 28: Within | 118 | 65 | 62 | 126 | 126 | 62 | 60 | 122
  WBC, Day 28: Above | 3 | 0 | 1 | 3 | 1 | 2 | 1 | 4
  WBC, Day 42: number analyzed (Participants) | 128 | 65 | 63 | 130 | 129 | 65 | 63 | 130
  WBC, Day 42: Unknown | 3 | 2 | 2 | 0 | 2 | 1 | 0 | 2
  WBC, Day 42: Below | 3 | 1 | 2 | 1 | 4 | 1 | 1 | 2
  WBC, Day 42: Within | 118 | 61 | 59 | 126 | 123 | 62 | 61 | 123
  WBC, Day 42: Above | 4 | 1 | 0 | 3 | 0 | 1 | 1 | 3
  WBC, Day 182: number analyzed (Participants) | 126 | 63 | 63 | 129 | 129 | 65 | 63 | 130
  WBC, Day 182: Unknown | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  WBC, Day 182: Below | 4 | 0 | 1 | 4 | 3 | 2 | 1 | 1
  WBC, Day 182: Within | 120 | 62 | 60 | 122 | 126 | 62 | 61 | 129
  WBC, Day 182: Above | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 0

42. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as the occurrence of any MAE regardless of intensity grade or relation to vaccination. Results were tabulated for subjects aged between 18 and 64 years and older (>64y).
Time Frame: Days 0 to 385
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 131 | 65 | 64 | 130
Participants
  Any MAEs, 18-64y: number analyzed (Participants) | 93 | 48 | 47 | 91 | 92 | 50 | 47 | 92
  Any MAEs, 18-64y | 49 | 24 | 14 | 32 | 38 | 23 | 23 | 36
  Any MAEs, >64y | 60 | 37 | 39 | 67 | 62 | 35 | 40 | 59

43. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Results were tabulated for subjects aged between 18-64 years and above 65 years (+65y).
Time Frame: Days 0 to 365
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 131 | 65 | 64 | 130
Participants
  Any pIMDs, 18-64y: number analyzed (Participants) | 93 | 48 | 47 | 91 | 92 | 50 | 47 | 92
  Any pIMDs, 18-64y | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any pIMDs, + 65y | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0

44. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 42-day (Days 0-41) post-vaccination period
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 222 | 114 | 112 | 221 | 223 | 115 | 111 | 222
Participants | 97 | 55 | 38 | 93 | 82 | 43 | 55 | 86

45. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Results were tabulated for subjects aged between 18-64 years and older (>64y).
Time Frame: Within the 84-day (Days 0-83) post-vaccination period
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 131 | 65 | 64 | 130
Participants
  Any AE(s), 18-64y: number analyzed (Participants) | 93 | 48 | 47 | 91 | 92 | 50 | 47 | 92
  Any AE(s), 18-64y | 51 | 29 | 18 | 46 | 36 | 26 | 27 | 44
  Any AE(s), > 64y | 66 | 32 | 32 | 62 | 61 | 30 | 35 | 64

46. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Results were tabulated for subjects aged between 18-64 years and older (>64y).
Time Frame: During the entire study period (from Day 0 to Day 385)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
Number analyzed (Participants) | 129 | 66 | 65 | 130 | 131 | 65 | 64 | 130
Participants
  Any SAE(s), 18-64y: number analyzed (Participants) | 93 | 48 | 47 | 91 | 92 | 50 | 47 | 92
  Any SAE(s), 18-64y | 7 | 0 | 2 | 1 | 2 | 1 | 2 | 3
  Any SAE(s), > 64y | 12 | 5 | 4 | 7 | 6 | 4 | 7 | 8

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) period post vaccine/placebo administration. Unsolicited AEs: during the 184-day (Days 0-183) post vaccine/placebo administration. Serious Adverse events (SAE): from Day 0 to Day 385.
Arm/Group | GSK2340274A F1_2D Group | GSK2340274A F2_2D Group | GSK2340274A F2_1D Group | GSK2340274A F1_1D Group | GSK2340273A F1_1D Group | GSK2340273A F2_2D Group | GSK2340273A F2_1D Group | GSK2340273A F3_2D Group
All-Cause Mortality (participants affected / at risk) | 1/222 | 1/114 | 0/112 | 0/221 | 0/223 | 0/115 | 0/111 | 1/222
Serious Adverse Events (participants affected / at risk) | 19/222 | 5/114 | 6/112 | 8/221 | 8/223 | 5/115 | 9/111 | 11/222
Other Adverse Events (participants affected / at risk) | 189/222 | 86/114 | 79/112 | 188/221 | 126/223 | 74/115 | 76/111 | 130/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340274A F1_2D Group (N=222) | GSK2340274A F2_2D Group (N=114) | GSK2340274A F2_1D Group (N=112) | GSK2340274A F1_1D Group (N=221) | GSK2340273A F1_1D Group (N=223) | GSK2340273A F2_2D Group (N=115) | GSK2340273A F2_1D Group (N=111) | GSK2340273A F3_2D Group (N=222)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340274A F1_2D Group (N=222) | GSK2340274A F2_2D Group (N=114) | GSK2340274A F2_1D Group (N=112) | GSK2340274A F1_1D Group (N=221) | GSK2340273A F1_1D Group (N=223) | GSK2340273A F2_2D Group (N=115) | GSK2340273A F2_1D Group (N=111) | GSK2340273A F3_2D Group (N=222)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (63) | 26 (36) | 11 (15) | 35 (40) | 35 (46) | 11 (13) | 11 (16) | 24 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 4 (6) | 2 (2)
Chills (General disorders) | 34 (37) | 17 (22) | 4 (4) | 17 (18) | 22 (27) | 12 (13) | 7 (9) | 25 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 7 (7) | 6 (7) | 10 (10) | 11 (11) | 4 (4) | 5 (6) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0) | 6 (7) | 10 (12) | 1 (1) | 1 (2) | 6 (11)
Erythema (Skin and subcutaneous tissue disorders) | 22 (25) | 0 (0) | 3 (3) | 14 (14) | 2 (2) | 2 (2) | 2 (2) | 7 (7)
Fatigue (General disorders) | 75 (108) | 42 (55) | 15 (21) | 67 (84) | 58 (72) | 26 (34) | 31 (41) | 45 (61)
Headache (Nervous system disorders) | 81 (108) | 37 (48) | 27 (34) | 64 (80) | 60 (81) | 32 (46) | 34 (49) | 55 (77)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 23 (25) | 8 (9) | 2 (3) | 10 (10) | 19 (20) | 4 (4) | 9 (10) | 12 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 83 (117) | 40 (60) | 14 (17) | 67 (82) | 44 (57) | 24 (27) | 23 (26) | 34 (44)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 7 (8) | 3 (5) | 8 (8) | 10 (11) | 1 (1) | 2 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 9 (9) | 4 (5) | 3 (3) | 7 (7) | 15 (15) | 8 (8) | 5 (6) | 14 (15)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (6) | 1 (1) | 1 (1) | 8 (8) | 6 (6) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) | 6 (6) | 8 (8) | 14 (15) | 8 (11) | 7 (7) | 14 (15)
Pain (General disorders) | 168 (279) | 76 (128) | 57 (61) | 156 (173) | 48 (62) | 27 (30) | 25 (28) | 42 (47)
Pyrexia (General disorders) | 11 (11) | 3 (3) | 1 (1) | 6 (7) | 13 (14) | 3 (4) | 7 (7) | 7 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 9 (11) | 3 (3) | 9 (11) | 4 (4)
Swelling (General disorders) | 20 (25) | 8 (9) | 4 (5) | 20 (21) | 7 (7) | 2 (2) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 5 (5) | 5 (5) | 7 (7) | 3 (3) | 4 (5) | 5 (5) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.